| S | tatistical | Analy | vsis | Plan | <b>H8H</b> - | -CD- | LAHE |
|---|------------|-------|------|------|--------------|------|------|

A Phase I, Multicenter, Open-Label, Parallel-Group, Pharmacokinetic Single Dose Study of Oral Lasmiditan in Subjects with Normal and Impaired Hepatic Function

NCT03040479

Approval Date: 24-Oct-2017

# **16.1.9 Documentation of Statistical Methods**

16.1.9.1. Statistical analysis plan (SAP)

16.1.9.2 Documentation of statistical analysis –  $SAS^{\mathbb{R}}$  output

Clinical Study Report Project N° COL MIG-114/H8H-CD-LAHF

# 16.1.9.1. Statistical analysis plan (SAP)

The statistical analysis plan (SAP) is presented next.



# STATISTICAL ANALYSIS PLAN

For:

CoLucid Pharmaceuticals, Inc.

SPONSOR PROTOCOL No. COL MIG-114

A Phase I, Multicenter, Open-Label, Parallel-Group, Pharmacokinetic Single Dose Study of Oral Lasmiditan in Subjects with Normal and Impaired Hepatic Function

Algorithme Project No. CUD-P9-453

Prepared by:

Algorithme Pharma 575 Armand-Frappier Laval, Quebec Canada, H7V 4B3

Version: Final 1.0

Date: 2017/10/24



# STATISTICAL ANALYSIS PLAN APPROVAL

We have carefully read this Statistical Analysis Plan and agree it contains the necessary information required to handle the statistical analysis of study data.

| PPD | |
|--------------------------|--------------------|
| PPD | 2017/11103<br>Date |
| On behalf of the Sponsor | Date |



# **VERSION CONTROL**

| Version<br>Number | Version Date | Author | Description of Significant Changes from Previous Approved Version |
|---|---|---|---|
| DRAFT 0.1 | 2017/08/11 | PPD<br>PPD | Not Applicable – First Version |
| DRAFT 0.2 | 2017/09/29 | PPD<br>PPD | Not Applicable – Second Version after the first round of comments |
| DRAFT 0.3 | 2017/10/16 | PPD<br>PPD | Not Applicable – Third Version after the second round of comments |
| DRAFT 0.4 | 2017/10/24 | PPD<br>PPD | Not Applicable – Fourth Version after the third round of comments |
| FINAL 1.0 | 2017/10/28 | PPD<br>PPD | / Final version |



# **CONTENTS**

| STATISTICAL ANALYSIS PLAN APPROVAL | 2 |
|-------------------------------------------------------|----------|
| VERSION CONTROL | 3 |
| ABBREVIATIONS | 6 |
| 1. INTRODUCTION | 7 |
| 2. STUDY OBJECTIVES | 8 |
| Primary Objectives | 8 |
| Secondary Objective | 8 |
| 3. STUDY DESIGN | 9 |
| General Description | 9 |
| Randomization and Unblinding Procedure | 9 |
| 4. STUDY ENDPOINTS | 10 |
| Pharmacokinetic Endpoints | 10 |
| Safety Endpoints | 10 |
| Sample Size Determination | 10 |
| 5. ANALYSIS POPULATIONS | 11 |
| 6. STATISTICAL METHODOLOGY | 12 |
| Analysis Time Points | 12 |
| Methods for Handling Missing Data | 12 |
| 7. STUDY SUBJECTS | 13 |
| Disposition Protocol Devictions | 13 |
| Protocol Deviations | 13 |
| 8. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 14 |
| Demographic and Background Characteristics Lifestyle | 14<br>14 |
| Medical/Social history | 14 |
| Prior Medication | 14 |
| 9. PHARMACOKINETICS AND STATISTICS | 15 |
| Pharmacokinetic Analysis | 15 |
| Statistical Analysis | 15 |
| 10. SAFETY | 17 |
| Adverse Events | 17 |
| Concomitant Medications | 17 |
| Extent of Exposure | 17<br>18 |
| Clinical Laboratory Evaluations Vital Signs | 18 |
| Electrocardiogram | 18 |
| Physical Examination Findings | 18 |
| Columbia-Suicide Severity Rating Scale (C-SSRS) | 18 |
| 11. INTERIM ANALYSES AND DATA SAFETY MONITORING | 19 |
| 12. CHANGES TO PROTOCOL-SPECIFIED ANALYSES | 20 |
| 13. GENERAL INFORMATION RELATED TO DATA PRESENTATIONS | 21 |
| PLANNED TABLES | 23 |



| PLANNED LISTINGS | 28 |
|---|---|
| APPENDIX A | 26 |
| APPENDIX B Pharmacokinetic Parameters | 27<br>27 |
| APPENDIX C TABLE SHELLS | 28<br>28 |
| APPENDIX D PHARMACOKINETIC OUTPUTS SHELLS PHARMACOKINETIC FIGURES SHELLS | 42<br>42<br>49 |
| APPENDIX E LISTING SHELLS | 55<br>58 |



## **ABBREVIATIONS**

AE Adverse Event

ANOVA Analysis of Variance

ATC Anatomical/Therapeutic/Chemical

AUC Area Under Curve
BMI Body Mass Index
CI Confidence Interval
CLCR Creatinine Clearance
CNS Central Nervous System
CRF Case Report Form
CS Clinically Significant

C-SSRS Columbia-Suicide Severity Rating Scale

CSR Clinical Study Report

eGRF Estimated Glomerular Filtration Rate

EOS End of Study

ICF Informed Consent Form

MedDRA Medical Dictionary for Regulatory Activities

NCS Not Clinically Significant
PK Pharmacokinetic(s)
SAE Serious Adverse Event
SAP Statistical Analysis Plan
SD Standard Deviation
SE Standard Error
SOC System Organ Class

TEAE Treatment-Emergent Adverse Event

TFLs Tables, Figures, and Listings
WHO-DDE WHO Drug Dictionary Enhanced



## 1. INTRODUCTION

This statistical analysis plan (SAP) provides a detailed description of the statistical methods and procedures to be implemented for the analyses of data from Protocol No. COL MIG-114. The analyses described in the SAP are based upon the final protocol (Fully signed) dated 2017/01/09.



## 2. STUDY OBJECTIVES

# Primary Objectives

The primary objective of this study is to evaluate the pharmacokinetic profile of lasmiditan following a single oral 200 mg dose in subjects with mild and moderate hepatic function relative to matched, healthy controls with normal hepatic function.

# Secondary Objective

The secondary objective of this study is to assess the safety and tolerability of a single oral 200 mg dose of lasmiditan in subjects with normal, mild and moderate hepatic function.



## 3. STUDY DESIGN

## General Description

This is a multi-center, open-label, non-randomized, parallel-group, single dose study. This study will enroll up to 24 subjects and will include 2 hepatic impaired subject groups and one group of control subjects with normal hepatic function.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered in the study.

Approximately four subjects with mild hepatic impairment will be enrolled first (Group 1). To ensure subject safety, following dosing of these first four subjects, a safety meeting will take place to review the safety data prior to dosing additional subjects. After safety and PK results from the first four subjects have been reviewed, an additional four subjects with mild hepatic impairment (remainder of Group 1) will be enrolled concurrently with the moderated hepatic impairment group (Group 2). Thereafter, matched subjects with normal hepatic function (Group 3) will be enrolled. There will be up to 8 subjects in each of the following groups, based on hepatic function at screening:

- Group 1: Mild hepatic impairment subjects (Child-Pugh Class A: 5 to 6 points)
- Group 2: Moderate hepatic impairment subjects (Child-Pugh Class B: 7 to 9 points)
- Group 3: Healthy subjects with normal hepatic function

All subjects will participate in one treatment period and will receive a single dose of lasmiditan in the fasting state. Subjects will be confined to the clinic from at least 10 hours prior to dosing until 36 hours after drug administration. The total duration of each subject's participation in the study will be 3 days (Day –1 through the last PK sample taken on Day 2), not including the screening and follow-up phone call. Study procedures

For complete details on the study assessments to be performed for the study, refer to Appendix A.

## Randomization and Unblinding Procedure

No randomization will be performed for this study No unblinding procedure is required, as this in an open-label study.



## 4. STUDY ENDPOINTS

## Pharmacokinetic Endpoints

The following plasma PK parameters of lasmiditan will be calculated:  $C_{max}$ ,  $T_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ , %AUC( $t_{last}$ - $\infty$ ),  $\lambda_z$ ,  $T_{1/2}$ , CL/F,  $V_z/F$ .

## Safety Endpoints

Safety endpoints include:

- Adverse Events
- Clinical Laboratory Tests (hematology, chemistry, urinalysis)
- Vital Signs
- Physical examination
- Concomitant medication
- 12 Lead ECGs
- C-SSRS

The details of the safety endpoints' assessment are presented in Section 10.

## Sample Size Determination

There is no formal statistical sample size calculation for this study. A sample size of 24; including 8 subjects/patients for each hepatic function group (8 subjects with normal hepatic function, 8 patients with mildly impaired hepatic function and 8 patients with moderately impaired hepatic function) was chosen because it is considered typical for studies evaluating the effect of hepatic function on the pharmacokinetics of a drug.



## 5. ANALYSIS POPULATIONS

#### **Safety Population:**

All subjects who received a dose of study medication will be included in the safety population. This population will be used for all demography and safety analyses.

### Pharmacokinetics (PK) Population:

All subjects who received lasmiditan, had no major protocol deviations, and completed the period with evaluable (sufficient and interpretable) data will be included in the PK population.

If some subjects do not complete the sampling schedule resulting in an inadequately characterized some PK parameters (e.g. AUC,  $V_Z/F$ ,  $\lambda_Z$ ), samples of these subjects could be included in the statistical pharmacokinetic analysis for only the evaluable parameters



## STATISTICAL METHODOLOGY

All analyses will be conducted using the SAS software, version 9.4, or higher. Descriptive statistics of the PK data will be performed by Phoenix® WinNonlin® version 6.3 or higher, Phoenix® ConnectTM version 1.3.1 or higher).

Adverse events and medical history will be classified using the standard MedDRA terminology version 19.1.

Prior and concomitant medications will be coded with the WHO-DDE dictionary version March 01, 2016.

In general, all summary tables will be presented for safety population. Summaries will be presented by hepatic function group.

In general, the data listings will include all enrolled subjects up to the point of study completion or discontinuation; exceptions will be listings pertaining to a subset of subjects only (e.g., subjects with blood sampling time deviations) or a subset of records/events (e.g., abnormal laboratory values).

Categorical variables will be summarized using the PROC FREQ procedure. Continuous variables will be summarized using the PROC UNIVARIATE procedure. For log-transformed endpoints, geometric mean, and coefficient of variation will also be presented.

The following general comments also apply to all statistical analyses and data presentations:

- Duration variables in days will be calculated using the general formula: (end date start date) +1.
- Individual subject listings of all data represented on the CRFs will be provided to facilitate the investigation of tabulated values and to allow for the clinical review of all efficacy and safety parameters.
- When assessments are repeated for a given timepoint, only the result which is closes to the dosing time will be included in the summary tables.

The analyses described in this plan are considered a priori, that they have been defined prior to database lock. Any analyses performed subsequent to database lock will be considered post hoc and exploratory. Post hoc analyses will be labeled as such in the corresponding statistical output and identified in the CSR.

#### **Analysis Time Points**

Unless otherwise specified, the baseline value will be defined as the last non-missing evaluation prior to the first dose of study medication.

#### Methods for Handling Missing Data

No imputations of values for missing data will be performed. All data recorded on the case report form will be included in the listings that will accompany the clinical study report.



## 7. STUDY SUBJECTS

## Disposition

The subject disposition will be summarized for all subjects enrolled in this study, including:

- The number of subjects enrolled;
- The number of screen failure subjects;
- The number of subjects screened;
- The number and percentage of subjects who completed the study;
- The number and percentage of subjects discontinued from the study by primary reason for discontinuation and overall;
- The number and percentage of subjects included in each of the safety and PK populations.

The percentages will be calculated using the number of subjects randomized as denominator.

A listing of subject's disposition will be provided. A listing of subjects included in each of the analysis populations will also be provided. Screen failure subjects will also be presented in a listing.

#### **Protocol Deviations**

Inclusion/exclusion criteria violations will be presented in a listing.

All deviations from the scheduled PK sampling time of 2 minutes or more for post dose samples will be taken into consideration for the evaluation of PK parameters.



## 8. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

## Demographic and Background Characteristics

Demographic data and baseline characteristics will be presented in a data listing and summarized by hepatic function group in a table. Quantitative assessments to be summarized are age, height, body weight and body mass index (BMI) at screening. Subject demographics include sex, age, ethnicity, race and country. Baseline characteristics include height, weight, and BMI.

## Lifestyle

Alcohol and smoking intake history will be recorded and presented in separate listings.

## Medical/Social history

Any medical history findings will be recorded and presented in a listing. The listing will include the coding terms (e.g., SOC and Preferred Term).

#### Prior Medication

Any medications taken including prescription, nonprescription, OTC (cold and antacid medications), dietary supplements, vitamins or herbal medications from screening to the first dose of the study drug will be recorded and presented as prior medications in a listing. The listing will include the coding terms (e.g., ATC and Preferred Term).



## PHARMACOKINETICS AND STATISTICS

## Pharmacokinetic Analysis

The PK parameters are presented in Section 4 and Appendix B. All reported sampling time deviations (see Section 7) will be taken into consideration for evaluation of plasma PK parameters.

Only quantifiable concentrations will be used to calculate PK parameters. An exception to this rule is made for concentrations below the quantification limit (BQL), which will be set to zero when all of the following conditions are met:

The time points occur before the first quantifiable concentration. All other BQL concentrations will be treated as missing sample.

The pharmacokinetic parameters will be estimated using a non-compartmental approach with a log-linear terminal phase assumption. The trapezoidal rule will be used to estimate the area under the curve, and the terminal phase will be estimated by maximizing the coefficient of determination estimated from the log-linear regression model. These parameters ( $AUC_{(0-\infty)}$ , %AUC(tlast- $\infty$ ),  $\lambda_Z$ ,  $T_{1/Z}$ , CL/F and Vz/F) will be estimated for individual concentration-time profiles only when the terminal log-linear phase cannot be reliably characterized using the following criteria:

- Phoenix® WinNonlin® Best fit range selection:
- R2 of at least 80%

In the case where less than 3 consecutive measurable plasma concentrations of lasmiditan are observed, the AUC parameters will not be estimated.

Additional pharmacokinetic parameters may be calculated if deemed appropriate.

Pharmacokinetic analyses and associated descriptive statistics will be generated using Phoenix® WinNonlin® Version 6.3 (or higher).

## Statistical Analysis

The natural logarithmic transformation of  $C_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ ,  $\lambda_Z$ , CL/F and  $V_Z/F$  will be used for all statistical inference.

Statistical analyses will be generated using validated SAS® (version 9.4 or higher) using the Reg (and Mixed, if applicable) procedure(s).

#### **Regression Analysis**

The Child-Pugh classification at baseline will be used as the primary measure of hepatic function for a regression analysis to evaluate the relationships between estimated hepatic function and PK parameters. Hepatic function in affected subjects will be entered in separate regression models as the following:

- Individual Child-Pugh scores;
- Hepatic Impairment Group:
  - 1. Child-Pugh classification A;
  - 2. Child-Pugh classification B;
  - 3. Subject with normal hepatic function

For each PK parameter except  $T_{max}$ , a regression analysis will be performed to assess the impact of impaired Hepatic Function, using a regression model of the form  $\alpha + \beta^*$  (Hepatic Function) +  $\epsilon$  where the errors ( $\epsilon$ ) will be assumed to be independent and normally distributed with mean zero and variance  $\sigma$ 2. The parameter  $\beta$  represents the correlation between the relevant PK parameter and the Hepatic Function which will be treated as a continuous variable.

Non-parametric methods based on the Wilcoxon rank sum test will be used to analyze differences in  $T_{max}$  between Hepatic Impairment Groups. The rank-transformed  $T_{max}$  will be used as the dependent variable in a regression model to analyze the relationship between Individual Child-Pugh score and  $T_{max}$ .



The following is the SAS code for the regression model including the individual Child-Pugh scores as Hepatic Function:

```
Proc Reg;
   Model PKparam = HepaticFunction;
Run;
```

Where HepaticFunction is individual Child-Pugh scores and PKparam is the value of the non-log-transformed or log transformed PK parameter.

The following is the SAS code for the regression model including the Hepatic Impairment Group as Hepatic Function:

```
Proc Reg;
   Model PKparam = GrpA GrpB;
Run;
```

Where HepaticFunction is Individual Child-Pugh scores in the first regression model and Hepatic Impairment Group in the second regression model and PKparam is the value of the non-log-transformed or log transformed PK parameter.

The hypothesis of the slope of trend being different from zero will be assumed if the two-sided test of the nullity of the parameter  $\beta$  is statistically significant at the 5% level.

#### **Analysis of Variance**

The effect on the pharmacokinetic parameters of the hepatic function will be done including the measurement of the hepatic function and using an analysis of variance (ANOVA). The ANOVA model will include the 3 groups of subjects (2 Child-Pugh classification groups and healthy volunteers) entered as fixed effects.

Pairwise comparisons of the 3 groups will be generated using the Tukey-Kramer's procedure of adjustment for multiple comparisons and statistical significance will be assessed at the two-sided 5% level. Heterogeneity of variance among groups will be assumed. Individual contrasts as well as the corresponding 90% confidence interval comparing each group will be computed.

```
Proc Mixed;
   Class FunctionGroup;
   Model PKparam = FunctionGroup;
   Repeated / Group = FunctionGroup;
   LSmeans FunctionGroup/ Pdiff=All CL Alpha=0.1 Adjust=Tukey;
Run;
```

Where FunctionGroup is the Hepatic Impairment Group and PKparam is the value of the non-log-transformed  $C_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$  or the log transformed  $C_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ .

Non-parametric methods will be used to analyze differences in  $T_{max}$  between the Mild and Moderate groups and the Normal group. In addition to the group-specific medians and ranges, the Hodges-Lehmann median, 90% CIs and p-values for the difference based on the Wilcoxon rank sum test statistic will be presented.



## 10. SAFETY

#### Adverse Events

An AE is defined as any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.

A suspected adverse reaction is any adverse event for which there is a reasonable possibility that the drug caused the adverse event. 'Reasonable possibility' means there is evidence to suggest a causal relationship between the drug and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

AEs occurring after the initiation of the treatment are referred to as treatment emergent adverse events (TEAEs).

As an overall summary of AEs, the following will be presented by hepatic function group and overall:

- Number of reported AEs;
- Number of reported TEAEs;
- Number and percentage of subjects experiencing TEAEs;
- Number and percentage of subjects experiencing a drug-related TEAE (i.e. those with a relationship classified as reasonable possibility)
- Number and percentage of TEAEs by relationship to study treatment (i.e. reasonable possibility);
- Number and percentage of TEAEs by severity;
- Number of reported SAEs (serious adverse events);
- Number and percentage of subjects experiencing SAEs;
- Number and percentage of subjects experiencing drug-related SAEs;
- Number and percentage of TEAEs leading to withdrawal; and
- SAEs with an outcome of death.

Frequency tables will be presented hepatic function group, system organ class and preferred term that summarize all Treatment Emergent Adverse Events (TEAEs) and all drug-related TEAEs.

Subject listings of all Adverse Events (AEs) including severity and relationship to study drug will be provided. AEs leading to withdrawal and SAEs will also be presented in separate listings.

#### Concomitant Medications

Medications taken after the first dose of study drug until after discharge from the study will be recorded. Concomitant medications will be presented in a listing. The medication name, active ingredient, dose, units, formulation, route, indication or reason taken, code, date and time taken will be presented. The listing will also include the coding terms (e.g., ATC and Preferred Term).

## Extent of Exposure

Details of drug dosing (actual treatment received, actual date and time of administration, dose administered, and route of administration) will be listed by subject.



## Clinical Laboratory Evaluations

Planned laboratory analyses include:

- General Biochemistry: Sodium, potassium, chloride, glucose, blood urea nitrogen (BUN), creatinine, CICr, eGFR, total bilirubin, alkaline phosphatase, Uric Acid at screening, AST, ALT and albumin;
- Hematology: White cell count with differential (absolute values of neutrophil, lymphocyte, monocyte, eosinophil, and basophil), red cell count, hemoglobin, hemoglobin A1c, hematocrit, mean corpuscular volume (MCV), and platelets count;
- Urinalysis: Color, appearance, specific gravity, pH, leukocyte, protein, glucose, ketones, bilirubin, blood, nitrite, urobilinogen. Microscopic examination will only be performed if the dipstick test is outside of the reference range for leukocyte, blood, nitrite or protein
- Other: serology, Endocrinology, urine drug screen and serum pregnancy.

Hematology, chemistry and quantitative urinalysis laboratory test results will be summarized by hepatic function group, parameter and visit and will also be presented in a listing

Separate listings of for serology, Endocrinology, urine drug screen and serum pregnancy will also be provided.

Subject listings of abnormal on-study laboratory values will be provided. Similarly, clinically significant on-study laboratory data will be presented in a second listing.

## Vital Signs

Vital signs will include the measurement of blood pressure, pulse rate, body temperature, and orthostatic blood pressure.

For all vital signs, raw values, at each time point will be summarized by hepatic function group, parameter and visit. Vital signs data will also be presented in a listing.

Subject listing of abnormal on-study vital signs values (Out-of-Range – Not Clinically Significant (NCS) or Clinically Significant (CS)) will be provided. Similarly, CS on-study vital signs values (Out-of-Range – CS) will be presented in a second listing.

## Electrocardiogram

A 12-lead ECG will be obtained throughout the study. In some cases, repeat abnormal ECGs may be obtained.

Raw values at each time point will be summarized by hepatic function group, parameter and visit and will also be presented in a listing. Overall safety assessment will also be presented in the listing.

A subject listing of abnormal on-study ECG assessments (Abnormal – NCS or Abnormal – CS) will be provided. Similarly, CS on-study ECG assessments (Abnormal – CS) will be presented in a second listing.

#### Physical Examination Findings

A physical examination will be conducted and will be presented in a listing.

### Columbia-Suicide Severity Rating Scale (C-SSRS)

The Columbia-Suicide Severity Rating Scale (C-SSRS) is a suicidal ideation rating scale. The scale identifies behaviors and thoughts that are associated with an increased risk of suicidal actions in the future.

Subjects who answer 'Yes' to any of the questions on the C-SSRS questionnaire will be presented in a listing.



## 11. INTERIM ANALYSES AND DATA SAFETY MONITORING

Approximately four subjects with mild hepatic impairment will be enrolled first (Group 1). To ensure subject safety, following dosing of these first four subjects, a safety meeting will take place to review the safety data prior to dosing additional subjects. After safety and PK results from the first four subjects have been reviewed, an additional four subjects with mild hepatic impairment (remainder of Group 1) will be enrolled concurrently with the moderated hepatic impairment group (Group 2). Thereafter, matched subjects with normal hepatic function (Group 3) will be enrolled.



# 12. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

There is no change from the planned analysis described in the protocol.



## 13. GENERAL INFORMATION RELATED TO DATA PRESENTATIONS

## Safety

All programs used to generate statistical analyses will be validated according to Algorithme Pharma's standard operating procedures.

TFLs will be displayed on letter size paper, 8 ½ inches by 11 inches, using the Courier New font.

In general, summary statistics for raw variables (i.e., variables measured at the study site or central laboratory) will be displayed as follows: if required minima, maxima, means, quartiles, standard deviations and confidence limits will be displayed to the same number of decimal places as the raw data; if required medians will be displayed to one additional decimal place.

Percentages will be displayed to one decimal place. Percentages between 0 and 0.1 (exclusive) will be displayed as '<0.1'. P-values will be displayed to 3 decimal places. P-values that are less than 0.001 will be displayed as '<0.001'.

The numbers of decimal places for summary statistics of derived variables (i.e., variables that are not measured by the study site but are calculated for analysis based on other measured variables) will be determined on a case by case basis. In general, minima and maxima will be displayed to the commonly used unit of precision for the parameter. Means, medians, quartiles, and confidence limits will be displayed to one additional decimal place and standard deviations will be displayed to two additional decimal places.

The formats and layouts of TFLs are provided in subsequent sections. Actual formats and layouts may be altered slightly from those presented in the templates as necessary to accommodate actual data or statistics. Minor format changes will not require updates to the SAP.

The tables and listings listed below are common data displays. Their numbering and general content follow the ICH E3 guidelines. Some of the tables and listings may not be applicable/appropriate/necessary for a particular study. Additional tables and listings may be included, provided the numbering scheme remains consistent with ICH E3.

#### PK Data

All programs used to generate statistical analyses will be validated according to Algorithme Pharma's standard operating procedures.

TFLs will be displayed on letter size paper, 8 ½ inches by 11 inches, using the Courier New font.

Raw variables (i.e., variables measured at the study site or central laboratory) will be displayed with the same number of decimal places as received as per bioanalytical laboratory. Derived variables (i.e., variables that are not measured by the study site but are calculated for analysis based on other measured variables) will be displayed as follow:

- All calculated pharmacokinetic parameter values should be reported to three significant digits.
- Observed concentration data, e.g. C<sub>max</sub>, should be reported as received.
- Observed time data, e.g. T<sub>max</sub>, should be reported as received.
- N should be reported as whole numbers
- Percentage values should be reported with whole numbers, except for the %AUC(tlast-∞).
- Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

Summary statistics of raw variables: minima, mean, geometric mean, median, maxima, and standard deviation, coefficient of variation will be displayed with the same number of decimal places as the raw data;



- The following summary statistics will be listed for all variables except T<sub>max</sub> and T<sub>1/2</sub>, arithmetic mean, SD, and CV; geometric mean and CV; N, minimum, maximum, and median.
- Summary statistics for T<sub>max</sub>, and other discrete parameters, will be limited to N, minimum, maximum, and median. Report not calculated (NC) for other statistics
- Summary statistics for T<sub>1/2</sub> will be limited to geometric mean and CV; N, minimum, maximum, and median. Report not calculated (NC) for other statistics.

Summary statistics of derived variables will be displayed with the same number of decimal places as the derived variable.



#### PLANNED TABLES

# **Demographic Data**

| Table 14.1.1 | Subject Disposition – All Subjects |
|---|---|
| Table 14.1.2.1 | Summary of Demographic Characteristics (Safety Population) |
| Table 14.1.2.2 | Summary of Demographic Characteristics (Pharmacokinetic Population) |

## **Pharmacokinetic Data**

| Table 14.2.1 | Statistical Analysis – SAS output |
|--------------|-----------------------------------|
|--------------|-----------------------------------|

## **Safety Data**

Tables in this section are based on the safety population unless otherwise stated.

| Table 14.3.1.1 | Summary of Adverse Events |
|---|---|
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term |
| Table 14.3.1.3 | Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term |
| Table 14.3.2.1 | Listing of Deaths, Other Serious and Significant Adverse Events |
| Table 14.3.2.2 | Listing of Treatment Emergent Adverse Events Leading to Withdrawal |
| Table 14.3.4.1 | Listing of Abnormal On-Study Laboratory Values |
| Table 14.3.4.2 | Listing of Clinically Significant On-Study Laboratory Values |
| Table 14.3.4.3 | Summary of Blood Chemistry |
| Table 14.3.4.4 | Summary of Hematology |
| Table 14.3.4.5 | Summary of Quantitative Urinalysis |
| Table 14.3.5.1 | Listing of Abnormal On-Study Vital Signs Values |
| Table 14.3.5.2 | Listing of Clinically Significant On-Study Vital Signs Values |
| Table 14.3.5.3 | Summary of Vital Signs |
| Table 14.3.6.1 | Listing of Abnormal On-Study ECG Assessments |
| Table 14.3.6.2 | Listing of Clinically Significant On-Study ECG Assessments |
| Table 14.3.6.3 | Summary of ECG Assessments |

## In text Tables:

PK Parameters of Lasmiditan

Summary of Statistical Analysis of Lasmiditan

## In text Figures:

Linear Profile of the Mean for Lasmiditan

Logarithmic Profile of the Mean for Lasmiditan

Linear Regression of In-Transformed  $C_{\text{max}}$  vs Child-Pugh scores

Linear Regression of In-Transformed  $AUC_{(0^{-\infty})}$  vs Child-Pugh scores

# In text Figures (Section 14):

Linear Regression of In-Transformed AUC<sub>(0-tlast)</sub> vs Child-Pugh scores



Appendix 16.2.6.1

Linear Regression of In-Transformed CL/F vs Child-Pugh scores

PK Tables – Plasma

| | T T T T T T T T T T T T T T T T T T T |
|---|---|
| | - Table X. Measured Human Plasma Concentrations |
| | - Table X. Cumulative Area Under the Curve |
| | <ul> <li>Table X. Pharmacokinetic Parameters X. Elimination Parameters</li> </ul> |
| | - Table X. Actual Sampling Time |
| Appendix 16.2.6.2 | PK – Figures |
| | - Figure x: Linear Profile of the Mean |
| | - Figure x: Logarithmic Profile of the Mean |
| | <ul> <li>Figure x: Individual Linear Profile of Subject x</li> </ul> |
| | - Figure x: Individual Logarithmic Profile of Subject |
| | - Figure x: Individual Elimination Profiles |



## PLANNED LISTINGS

| Listing 16.2.1 | Listing of Study Disposition |
|---|---|
| Listing 16.2.2.1 | Listing of PK Blood Sampling Time Deviations |
| Listing 16.2.2.2 | Listing of Protocol Deviations |
| Listing 16.2.3 | Listing of Analysis Populations |
| Listing 16.2.4.1 | Listing of Demographic Characteristics |
| Listing 16.2.4.2 | Listing of Screen Failure Subjects |
| Listing 16.2.5 | Listing of Investigational Product Administration |
| Listing 16.2.7 | Listing of Adverse Events |
| Listing 16.2.8.1 | Listing of Blood Chemistry |
| Listing 16.2.8.2 | Listing of Hematology |
| Listing 16.2.8.3 | Listing of Urinalysis |
| Listing 16.2.8.4 | Listing of Urine Drug Screen |
| Listing 16.2.8.5 | Listing of Pregnancy Test |
| Listing 16.2.8.6 | Listing of Serology |
| Listing 16.2.8.7 | Listing of Endocrinology |
| Listing 16.2.9.1 | Listing of Alcohol Habits |
| Listing 16.2.9.2 | Listing of Smoking Habits |
| Listing 16.2.9.3 | Listing of Prior Medication |
| Listing 16.2.9.4 | Listing of Concomitant Medication |
| Listing 16.2.9.5 | Listing of Physical Examination |
| Listing 16.2.9.6 | Listing of Vital Signs |
| Listing 16.2.9.7 | Listing of ECG Assessments |
| Listing 16.2.9.8 | Listing of Inclusion/Exclusion Criteria Summary |
| Listing 16.2.9.9 | Listing of Medical History |
| Listing 16.2.9.10 | Listing of Columbia-Suicide Severity Rating Scale (C-SSRS) |



## **APPENDIX A**

#### STUDY SCHEDULE

| Examination | Screening Days | | | | Post-<br>Study<br>Tests or<br>ET <sup>a</sup> | End of Study |
|---|---|---|---|---|---|---|
| | Day 28 to -1 | -1 | 1 | 2 | 2 | 7 (±3) |
| Review Inc/Exclusion Criteria &<br>MedicalHistory | X | | | | | |
| Informed Consent | X | | | | | |
| Check-in | | X | | | | |
| Dosing | | | X | | | |
| Clinic Confinement | | X | X | X | | |
| Discharge | | | | X | | |
| Demographics | X | | | | | |
| C-SSRS questionnaire | X | | | | X | |
| Concomitant Medication | X | X | X | X | X | X |
| Physical Examination | X | | | | X | |
| Vital Signs <sup>b</sup> | X | | X | | X | |
| Height, Weight, and BMI | X | | | | | |
| 12-lead ECG <sup>c</sup> | X | | X | | X | |
| HIV Ag/Ab Combo, HBsAg (B) (Hepatitis<br>B) and HCV (C) Tests | X | | | | | |
| Drug and Alcohol Screen | X | X | | | | |
| Pregnancy test (females) | X | X | | | X | |
| Clinical Laboratory Evaluations <sup>d</sup> | X | X | | | X | |
| PK Blood Sample <sup>e</sup> | | | X | X | | |
| Follow-up Call | | | | | | X |
| Adverse Events Recording | X | X | X | X | X | X |

a Early Termination (ET).

b Vital signs will be measured prior to dosing and approximately 2 and 4 hours after study drug administration.

c 12-lead ECG will be performed prior to dosing and approximately 2 hours after study drug administration.

d Clinical laboratory tests (hematology, biochemistry, endocrinology (screening only) and urinalysis) will be performed. On Day -1, these will be done in the evening prior to drug administration.

e PK blood and urine samples will be collected according to schedule of PK assessments



# **APPENDIX B**

## Pharmacokinetic Parameters

| PK Parameter | Definition |
|---|---|
| $C_{max}$ | Maximum observed plasma concentration |
| $T_{\text{max}}$ | Time of maximum observed plasma concentration; if it occurs at more than one time point, $T_{max}$ is defined as the first time point with this value |
| AUC <sub>(0-tlast)</sub> | Cumulative area under the plasma concentration time curve calculated from 0 to $T_{LQC}$ using the linear trapezoidal method, where $T_{LQC}$ represents time of last observed quantifiable plasma concentration |
| $\mathrm{AUC}_{(0\text{-}\infty)}$ | Area under the plasma concentration time curve extrapolated to infinity, calculated as $AUC_{(0\text{-tlast})} + \hat{C}_{LQC}/\lambda_Z$ , where $\hat{C}_{LQC}$ is the estimated concentration at time $T_{LQC}$ |
| %AUC(t <sub>last</sub> -∞) | Relative percentage of AUC <sub>(0-tlast)</sub> with respect to AUC <sub>(0-∞)</sub> $\% AUC(t_{last} - \infty) = 100 \times \frac{\left(AUC(0-\infty) - AUC(0-t_{last})\right)}{AUC(0-\infty)}$ |
| $\lambda_{\mathrm{Z}}$ | Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration <i>versus</i> time curve |
| $T_{1/2}$ | Terminal elimination half-life, calculated as $ln(2)/\lambda_Z$ |
| CL/F | Apparent Total Plasma Clearance, calculated as dose /AUC <sub>(0-∞)</sub> |
| $V_z/F$ | Apparent Volume of Distribution, calculated as dose / $\lambda_Z$ *AUC <sub>(0-<math>\infty</math>)</sub> |



# **APPENDIX C**

## TABLE SHELLS

CoLucid Pharmaceuticals, Inc.
Project # COL MIG-114/CUD-P9-453


Table 14.1.1
Subject Disposition
(All Subjects)

| | | Healthy<br>Hepatic<br>Function<br>(N=XX) | Mild<br>Hepatic<br>Function<br>(N=XX) | Moderate<br>Hepatic<br>Function<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Subjects Enrolled | | XX | XX | XX | XX |
| Screen Fail Subjects | | XX | XX | xx | xx |
| Subjects Screened [N] | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects Completed the Study [n(%)] | YES<br>NO | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| If No, Reason of Study Discontinuation $[n(%)]$ | Reason 1<br>Reason 2<br>Reason 3<br>Etc. | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Number of Subjects Included in Each Analysis Population $[n(%)]$ | Safety Population<br>Pharmacokinetic Population | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

Note: The percentages are based on the number of subjects screened.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas




# Table 14.1.2.1 Summary of Demographic Characteristics (Safety Population)

| | | Healthy Hepatic<br>Function<br>(N=XX) | Mild Hepatic<br>Function<br>(N=XX) | Moderate<br>Hepatic<br>Function<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Age (years) | N | XX | XX | XX | XX |
| 3- (2/ | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Gender [n(%)] | MALE<br>FEMALE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity [n(%)] | HISPANIC/LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | NOT HISPANIC/NOT LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race [n(%)] | RACE1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | RACE2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Weight (kg) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Height (cm) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Body Mass Index(kg/m²) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |

Date: VERSION - YYYY-MM-DD

Similar Table:

Data Source: XXXX

Program Source: XXXXX.sas

Table 14.1.2.2 Summary of Demographic Characteristics (Pharmacokinetic Population)




# Table 14.3.1.1 Summary of Adverse Events (Safety Population)

| | Healthy Hepatic<br>Function<br>(N=XX) | Mild Hepatic<br>Function<br>(N=XX) | Moderate<br>Hepatic<br>Function<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Adverse Events (AEs) Reported [n] | | | | XX |
| Treatment Emergent Adverse Events (TEAEs) Reported [n] | XX | XX | XX | XX |
| Subjects With At Least One TEAE [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects With At Least One Drug-Related TEAE $[n(%)]$ [1] [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Relationship [2] Related [n(%)] [3] Not Related [n(%)] | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| <pre>TEAEs Severity/Intensity [2] Mild [n(%)] Moderate [n(%)] Severe [n(%)] Life-Threatening [n(%)]</pre> | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Serious Adverse Events (SAEs) Reported [n] [2] | XX | XX | XX | XX |
| Subjects With At Least One SAE [n(%)][1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject With an TEAE Leading to Withdrawal [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> Percentages are based on the number of subjects in the Safety population in each treatment group.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

<sup>[2]</sup> Percentages are based on the total number of treatment emergent adverse events reported in each treatment group.

<sup>[3]</sup> TEAE that was reported with a relationship of "reasonable possibility".




| SOC<br>MedDRA Preferred Term | Healthy Hepatic<br>Function<br>(N=XX) | Mild Hepatic Function (N=XX) | Moderate Hepatic Function (N=XX) |
|---|---|---|---|
| Subjects With At Least One TEAE [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MedDRA Term 11 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MedDRA Term 12 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MedDRA Term 13 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MedDRA Term 21 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MedDRA Term 22 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MedDRA Term 23 [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Each treatment emergent adverse event is counted only once for each subject within each System Organ Class and MedDRA Preferred Term.

Date: VERSION - YYYY-MM-DD Data Source: XXXXX Program Source: XXXXX.sas

Similar Table: Table 14.3.1.3 Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term




# Table 14.3.2.1 Listing of Deaths, Other Serious and Significant Adverse Events (Safety Population)

| Subject ID | Visit/<br>Group/<br>AE # | SOC MedDRA Preferred Term Description of AE | Onset Date<br>Time<br>(Time since<br>Last Dose) | Resolution<br>Date Time<br>(Duration) | S: Severity<br>R: Relationship<br>to Study Drug | O: Outcome<br>S: Serious AE<br>D: AE Leading To<br>Discontinuation | |
|---|---|---|---|---|---|---|---|
| xxx | xxxxx<br>xxxxx | ************************************** | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | YYYY-MM-<br>DD/<br>HH:MM<br>(DD:HH:MM) | xxxxxx | xxxxx | xxxxxx |

#### Similar Tables:

14.3.2.2 Listing of Treatment Emergent Adverse Events Leading to Withdrawal




# Table 14.3.4.1 Listing of Abnormal On-Study Laboratory Values (Safety Population)

| Category/ | Reference | | | | | Out-of-Rand | Out-of-Range |
|---|---|---|---|---|---|---|---|
| Parameter (Unit) | Range | Subject ID | Visit | Date / Time | Value | Flag | Assessment [1] |
| Lab Category 1 | | | | | | | |
| Lab Test 11 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | xxx | XXX |
| Lab Test 12 | xxx-xxx | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Lab Category 2 | | | | | | | |
| Lab Test 21 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Lab Test 22 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Etc. | xxx-xxx | XXX | XXXXXX | XXXXXX | XXX | xxx | XXX |

[1] NCS: Not Clinically Significant / CS: Clinically Significant / TBC: To Be Controlled.

Note(s): Abnormal values are determined by applying the reference ranges to the results as reported by the external laboratory analysis.

Date: VERSION - YYYY-MM-DD Data Source: XXXXX Program Source: XXXXX.sas



## Table 14.3.4.2 Listing of Clinically Significant On-Study Laboratory Values (Safety Population)

| Category/<br>Parameter (Unit) | Reference Range | Subject ID | Visit | Date / Time | Value | Out-of-<br>Range Flag | Assessment [1] |
|---|---|---|---|---|---|---|---|
| Lab Category 1<br>Lab Test 11 | xxx-xxx | xxx | xxxxxx | xxxxxx | xxx | xxx | xxx |
| Lab Test 12 | xxx-xxx | XXX | xxxxxx | XXXXXX | XXX | XXX | xxx |
| Lab Category 2<br>Lab Test 21 | xxx-xxx | xxx | xxxxxx | xxxxxx | xxx | xxx | xxx |
| Lab Test 22 | xxx-xxx | xxx | XXXXXX | xxxxxx | xxx | XXX | xxx |
| Etc. | xxx-xxx | xxx | xxxxxx | xxxxxx | xxx | XXX | xxx |

[1] CS: Clinically Significant / TBC: To Be Controlled.

Note(s): Abnormal values are determined by applying the reference ranges to the results as reported by the external laboratory analysis.




#### Table 14.3.4.3 Summary of Blood Chemistry (Safety Population)

| Parameter (unit) | Visit Name | | Statistic | Healthy Hepatic<br>Function<br>(N=XX) | Mild Hepatic<br>Function<br>(N=XX) | Moderate Hepatic<br>Function<br>(N=XX) |
|---|---|---|---|---|---|---|
| xxx (xxx) | Screening | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| | Day -1 | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| | Etc. | | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Tables:

14.3.4.4 Summary of Hematology

14.3.4.5 Summary of Quantitative Urinalysis




# Table 14.3.5.1 Listing of Abnormal On-Study Vital Signs Values (Safety Population)

| Assessment (Units) | Subject ID | Visit | Position | Date / Time | Value | Safety Review |
|---|---|---|---|---|---|---|
| Vital Sign Test 1 | | | xxxxxx | YYYY-MM-DD:XX:XX | XXX | xxx |
| vicar bign rese i | XXX | XXXXXX | | YYYY-MM-DD:XX:XX | | |
| | XXX | XXXXXX | XXXXXX | YYYY-MM-DD;XX:XX | XXX | XXX |
| Vital Sign Test 2 | XXX | xxxxxx | xxxxxx | YYYY-MM-DD:XX:XX | XXX | xxx |
| | XXX | xxxxxx | XXXXXX | YYYY-MM-DD:XX:XX | XXX | xxx |
| Etc. | XXX | xxxxxx | XXXXXX | YYYY-MM-DD;XX;XX | XXX | XXX |




# Table 14.3.5.2 Listing of Clinically Significant On-Study Vital Signs Values (Safety Population)

| Assessment (Units) | Subject ID | Visit | Position | Date / Time | Value | Safety Review |
|---|---|---|---|---|---|---|
| Vital Sign Test 1 | XXX | XXXXXX | XXXXXX | YYYY-MM-DD:XX:XX | XXX | XXX |
| | XXX | XXXXXX | xxxxxx | YYYY-MM-DD:XX:XX | XXX | XXX |
| Vital Sign Test 2 | xxx | xxxxxx | XXXXXX | YYYY-MM-DD:XX:XX | XXX | xxx |
| | xxx | xxxxxx | XXXXXX | YYYY-MM-DD:XX:XX | XXX | xxx |
| Etc. | xxx | xxxxxx | XXXXXX | YYYY-MM-DD:XX:XX | XXX | xxx |




#### Table 14.3.5.3 Summary of Vital Signs (Safety Population)

| Parameter (unit) | Visit | Timepoint | E | Statistic | Healthy Hepatic<br>Function<br>(N=XX) | Mild Hepatic<br>Function<br>(N=XX) | Moderate<br>Hepatic<br>Function<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| Vital Sign Test 1 | Screening | | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day 1 | 2 Hours | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day 1 | 4 Hours | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| Etc. | Etc. | | | | | | |

PROGRAMMING NOTE: All visits outlined in Appendix A will be included.




# Table 14.3.6.1 Listing of Abnormal On-Study ECG Assessments (Safety Population)

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | XXXXXX |
| | XXXXXX | XXX | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxx | XXXXXX |
| xxxxx | xxxxxx | xxx | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| xxxxx | xxxxxx | xxx | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |




# Table 14.3.6.2 Listing of Clinically On-Study ECG Assessments (Safety Population)

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| XXXXX | XXXXXX | xxx<br>xxx | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx<br>xxxxxx |
| xxxxx | xxxxxx | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx |




## Table 14.3.6.3 Summary of ECG Assessments (Safety Population)

| Parameter (unit) | Visit | | | | Healthy Hepatic<br>Function<br>(N=XX) | Mild Hepatic<br>Function<br>(N=XX) | Moderate<br>Hepatic<br>Function |
|---|---|---|---|---|---|---|---|
| | | Timepoint | | Statistic | | | (N=XX) |
| ECG Assessment Test 1 | | | | | | | |
| | Screening | | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day -1 | | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day 1 | Pre-dose | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| Etc. | Etc. | | | | | | |



## **APPENDIX D**

## PHARMACOKINETIC OUTPUTS SHELLS

Measured Human Plasma Concentrations of Lasmiditan, Normal Hepatic Function, CUD-P9-453

| | | | | | | Time<br>(h) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | | <br> | <br> | 36.00 |
| Hepatic Function | Subject | | | | | ncentra<br>(ng/m | | | |
| Normal | 101 | | | | | | | | |
| | 108 | | | | | | | | |
| | N | | | | | | | | |
| | Mean | | | | | | | | |
| | SD | | | | | | | | |
| | Min | | | | | | | | |
| | Median | | | | | | | | |
| | Max | | | | | | | | |
| | CV% | | | | | | | | |
| | <b>Geometric Mean</b> | | | | | | | | |
| | Geometric CV% | | | | | | | | |
| | | BLQ: | Below Li | mit of Qua | antitation | 1 | | | |
| | | | NC: Not | Calculate | ed | | | | |



Similar tables will be presented for all hepatic groups



## Cumulative Area Under the Curve of Lasmiditan, Normal Hepatic Function, CUD-P9-453

| | | | | | | Time<br>(h) | |
|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | | 36.00 |
| Hepatic Function | Subject | Cumulative AUC<br>(ng*h/mL) | | | | | |
| Normal | 101 | | | | | | |
| | 108 | | | | | | |
| | N | | | | | | |
| | Mean | | | | | | |
| | SD | | | | | | |
| | Min | | | | | | |
| | Median | | | | | | |
| | Max | | | | | | |
| | CV% | | | | | | |
| | <b>Geometric Mean</b> | | | | | | |
| | Geometric CV% | | | | | | |
| | | | NC: Not | Calculate | ed | | |

Similar tables will be presented for all hepatic groups and for urine data by intervals.



## Pharmacokinetic Parameters of Lasmiditan, Normal Hepatic Function, CUD-P9-453

| Hepatic Function | Subject | C <sub>max</sub><br>(ng/mL) | T <sub>max</sub><br>(h) | AUC <sub>(0-Tlast)</sub><br>(ng*h/mL) | AUC <sub>(0-∞)</sub><br>(ng*h/mL) | %AUC <sub>(tlast-</sub><br>-∞) (%) | T <sub>1/2</sub> (h) | CL/F<br>(L/h) | V <sub>z</sub> /F<br>(L) |
|---|---|---|---|---|---|---|---|---|---|
| Normal | 101 | | | | | | | | |
| | 108 | | | | | | | | |
| | N | | | | | | | | |
| | Mean | | NC | | | | NC | | |
| | SD | | NC | | | | NC | | |
| | Min | | | | | | | | |
| | Median | | | | | | | | |
| | Max | | | | | | | | |
| | CV% | | NC | | | | NC | | |
| | <b>Geometric Mean</b> | | NC | | | | | | |
| 0: " + 11 " | Geometric CV% | 1, | NC | | | | | | |

Similar tables will be presented for all hepatic groups and for urine parameters.



## Elimination Parameters of Lasmiditan, Normal Hepatic Function, CUD-P9-453

| Hepatic Function | Subject | T <sub>LIN</sub> (h) | T <sub>LQC</sub> (h) | Number of Points | R <sup>2</sup> | λ <sub>z</sub><br>(1/h) |
|---|---|---|---|---|---|---|
| Normal | 101 | | | | | |
| | 108 | | | | | |
| | N | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Min | | | | | |
| | Median | | | | | |
| | Max | | | | | |
| | CV% | | | | | |
| | <b>Geometric Mean</b> | | | | | |
| | Geometric CV% | | | | | |

A similar table will be presented for all hepatic groups.



## Actual Sampling Time of Lasmiditan, Normal Hepatic Function, CUD-P9-453

| | | Time<br>(h) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | | | | | <br> | <br> | <br>36.00 |
| Hepatic Function | Subject | | 1 | | L | 1 | A | ctual Ti<br>(h) | me | | 1 | |
| Normal | 101 | | | | | | | | | | | |
| | ••• | | | | | | | | | | | |
| | 108 | | | | | | | | | | | |
| | N | | | | | | | | | | | |
| | Mean | | | | | | | | | | | |
| | SD | | | | | | | | | | | |
| | Min | | | | | | | | | | | |
| | Median | | | | | | | | | | | |
| | Max | | | | | | | | | | | |
| | CV% | | | | | | | | | | | |
| | Geometric Mean | | | | | | | | | | | |
| | Geometric CV% | | | | | | | | | | | |
| | | | | NC | : Not Cald | culated | | | | | | |

A similar table will be presented for all hepatic groups.



## Pairwise Comparisons of Lasmiditan, CUD-P9-453

| Parameters | Geometric LSmea | ns <sup>a</sup> Comparison | Adjusted p- | Ratio | 90% Confidence Limits (%) | |
|---|---|---|---|---|---|---|
| r drameters | Group | Companson | value | (%) | Lower | Upper |
| | Mild (n=x) | Mild vs Moderate | | | | |
| $C_{max}$ | Moderate (n=x) | Mild vs Normal | | | | |
| | Normal (n=x) | Moderate vs Normal | | | | |
| | Mild (n=x) | Mild vs Moderate | | | | |
| AUC <sub>(0-tlast)</sub> | Moderate (n=x) | Mild vs Normal | | | | |
| | Normal (n=x) | Moderate vs Normal | | | | |
| | Mild (n=x) | Mild vs Moderate | | | - | |
| $AUC_{(0-\infty)}$ | Moderate (n=x) | Mild vs Normal | | | | |
| | Normal (n=x) | Moderate vs Normal | | | | |

a C<sub>max</sub> is presented in ng/mL, AUC<sub>(0-tlast)</sub> and AUC<sub>(0-∞)</sub> are presented in ng\*h/mL

### Paired Comparisons of Tmax, Lasmiditan, CUD-P9-453

| | Median | (Range) | | P-value for | Hodges-<br>Lehmann<br>Median for | 90% Confidence Limits for<br>Difference from Control | |
|---|---|---|---|---|---|---|---|
| Parameter | Group | | Comparison | Difference | Difference<br>from Control | Lower | Upper |
| | Mild (n=x) | | Mild vs Moderate | | | | |
| $T_{max}$ | Moderate (n=x) | | Mild vs Normal | | | | |
| | Normal (n=x) | | Moderate vs Normal | | | | |

Tmax was analyzed using the Wilcoxon rank sum test



### PHARMACOKINETIC FIGURES SHELLS

Figure 1: Linear Profile of the Mean of Lasmiditan in Plasma





Figure 2: Logarithmic Profile of the Mean of Lasmiditan in Plasma





Figures 2+1 to (2+1)+N: Individual Linear Profile of Lasmiditan in Plasma

SubjectNumber=101, RenalGroup=Normal





Figure X: Individual Logarithmic Profile of Lasmiditan in Plasma

### SubjectNumber=101, RenalGroup=Normal





Figure N: Individual Elimination Profiles

SubjectNumber=101, Group=1, RenalGroup=Nomal R2=0.992 Rsq\_adjusted=0.9879 Thalf=5.0521 4 points used in calculation Uniform Weighting





In Text Figure:



The figure does not reflect the actual data of the study. Same graph will be presented for  $AUC_{(0-\text{tlast})}$ ,  $AUC_{(0-\infty)}$  and CL/F.



## **APPENDIX E**

LISTING SHELLS




#### Listing 16.2.1 Listing of Study Disposition

| | Date of Completion or | | | | |
|---|---|---|---|---|---|
| Subject ID | Discontinuation | Subject Status | Specify | AE # | Date of Death |




## Listing 16.2.2.1 Listing of PK Blood Sampling Time Deviations

| | Elapsed | | Scheduled | Actual | |
|-------|----------|------------|-----------|-----------|-----------------|
| Group | Time (h) | Subject ID | Date/Time | Date/Time | Deviation (min) |




#### Listing 16.2.3 Listing of Analysis Populations

| | Safety | |
|---|---|---|
| Subject ID | Population PK Population | Reason if Excluded from one Population |




## Listing 16.2.4.1 Listing of Demographic Characteristics

|--|




### Listing 16.2.4.2 Listing of Screen Failures

Subject ID Date Specify Primary Reason




#### Listing 16.2.5 Listing of Investigational Product Administration

| | | Start | | Dose | | If Any Dosi | ng Issues, |
|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Date/Time | Treatment | Administered (mg) | Route | Specify | |




#### Listing 16.2.7 Listing of Adverse Events

| Subject ID | Visit/<br>Group/<br>AE # | SOC MedDRA Preferred Term Description of AE | Onset Date<br>Time<br>(Time since<br>Last Dose) | Resolution<br>Date Time<br>(Duration) | S: Severity R: Relationship to Study Drug | O: Outcome S: Serious AE D: AE Leading To Discontinuation | Action Taken With Study Treatment / Other Action(s) Taken / Concomitant Given |
|---|---|---|---|---|---|---|---|
| xxx | xxxxx<br>xxxxx | ************************************** | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | xxxxx | xxxxx | xxxxxx |




#### Listing 16.2.8.1 Listing of Blood Chemistry

| | | | | | | | Out-of-Range | Assessment |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Lab Test Name (Units) | Reference Range | Visit | Date / | Time | Value | Flag | [1] |

[1] NCS: Not Clinically Significant / CS: Clinically Significant / TBC: To Be Controlled.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

### Similar listing(s):

| L16.2.8.2 | Listing | of | Hematology |
|-----------|---------|----|-------------------|
| L16.2.8.3 | Listing | of | Urinalysis |
| L16.2.8.4 | Listing | of | Urine Drug Screen |
| L16.2.8.5 | Listing | of | Pregnancy Test |
| L16.2.8.6 | Listing | of | Serology |
| L16.2.8.7 | Listing | of | Endocrinology |




#### Listing 16.2.9.1 Listing of Alcohol Habits

| Subject ID | Intake Status | Quantity | Frequency | Start Date | End Date |
|------------|---------------|----------|-----------|------------|----------|
|------------|---------------|----------|-----------|------------|----------|




#### Listing 16.2.9.2 Listing of Smoking Habits

| Subject ID Intake Status Quantity Frequency | Start Date End Date |
|---------------------------------------------|---------------------|
|---------------------------------------------|---------------------|




## Listing 16.2.9.3 Listing of Prior Medication

| | | | ATC / | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | PT / | | | | | Total | | Start | End |
| | | Related to | Medication | | Dose | | | Daily | | Date/ | Date/ |
| Subject ID | #CM | AE#/MH# | Name | Indication | (unit) | Frequency | Formulation | Dose | Route | Time | Time |

Date: VERSION - YYYY-MM-DD Data Source: XXXXX Program Source: XXXXX.sas

Similar Listing:

Listing 16.2.9.4 Listing of Concomitant Medication




## Listing 16.2.9.5 Listing of Physical Examination

| Subject ID | Visit | Date / Time | Body System Examined | Result | (Abnormal Findings) |
|---|---|---|---|---|---|




### Listing 16.2.9.6 Listing of Vital Signs

| | | | | | Assessment | Safety |
|---|---|---|---|---|---|---|
| Subject ID | Visit | Timepoint | Position | Date / Time | (Units) Val | ue Review |




#### Listing 16.2.9.7 Listing of ECG Assessments

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | | YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx |
| | | | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx<br>xxxxxx |
| XXXXX | XXXXX | | YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx |
| xxxxx | xxxxxx | | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |


CoLucid Pharmaceuticals, Inc.
Project # COL MIG-114/CUD-P9-453


# Listing 16.2.9.8 Listing of Inclusion/Exclusion Criteria Summary

Has the participant met all
Subject ID screening eligibility criteria? Inclusion/Exclusion Failed Criterion Number

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas



CoLucid Pharmaceuticals, Inc.
Project # COL MIG-114/CUD-P9-453


#### Listing 16.2.9.9 Listing of Medical History

| | | | Description of Medical | | |
|---|---|---|---|---|---|
| Subject ID | MH # System Organ Class | MedDRA Preferred Term | History | Start Date | End Date |

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas



CoLucid Pharmaceuticals, Inc.
Project # COL MIG-114/CUD-P9-453

CONFIDENTIAL
Page 1 of x

# Listing 16.2.9.10 Listing of Columbia-Suicide Severity Rating Scale (C-SSRS)

| Subject is vibit Subject on into the subject of the | Subject ID | Visit | Category | Question | Answer |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas



## contact@altasciences.com

<u>altasciences.com</u>



575 Armand-Frappier Blvd. Laval, Quebec Canada H7V 4B3 450 973-6077 algopharm.com



10103 Metcalf Ave.

Overland Park, KS 66212

United States
913 696-1601

vinceandassociates.com



4837 Amber Valley Parkway Fargo, ND 58104 United States 701 551-3737 algopharm.com

# 16.1.9.2 Documentation of statistical analysis – $SAS^{\circledR}$ output

Legend: AUCinf= AUC $_{0-\infty}$ 

$$\begin{split} AUCT &= AUC_{0\text{-Tlast}} \\ LambdaZ &= \lambda_Z \\ Vz\_F &= V_z/F \\ CL\_F &= CL/F \\ lCmax &= ln(C_{max}) \end{split}$$

$$\begin{split} &lAUCT = ln(AUC_{0\text{-Tlast}}) \\ &lAUCinf = ln(AUC_{0-\infty}) \end{split}$$

 $\begin{aligned} &\text{IVz}\_F = \ln(\text{V}_z/\text{F}) \\ &\text{ICL}\_F = \ln\left(\text{CL/F}\right) \\ &\text{RkTmax} = \text{Rank of T}_{\text{max}} \end{aligned}$ 

# RAW DATA

#### Hepatic Function Group=Mild

| | | | | He | epatic Funct | tion Group= | :M11d | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Subject<br>ID | Cmax | Tmax | AUCT | AUCinf | Vz_F | Cl_F | LambdaZ | log{Cmax} | log{AUCT} | |
| 1 | 01401 | 159.00000 | 2.00000 | 1229.31750 | 1261.85792 | 1586.25544 | 158.49645 | 0.09992 | 5.06890 | 7.11421 | |
| 2 | 01402 | 350.00000 | 0.75000 | 1629.60250 | 1673.31600 | 1370.20933 | 119.52315 | 0.08723 | 5.85793 | 7.39609 | |
| 3 | 01404 | 125.00000 | 2.00000 | 978.55250 | 1007.61169 | 1257.71336 | 198.48916 | 0.15782 | 4.82831 | 6.88607 | |
| 4 | 01408 | 518.00000 | 0.75000 | 2019.77500 | 2033.41542 | 507.28430 | 98.35668 | 0.19389 | 6.24998 | 7.61074 | |
| 5 | 04101 | 255.00000 | 2.50000 | 2212.32550 | 2264.40458 | 855.45252 | 88.32344 | 0.10325 | 5.54126 | 7.70180 | |
| 6 | 04102 | 258.00000 | 2.50000 | 1603.91250 | 1635.53001 | 744.38302 | 122.28452 | 0.16428 | 5.55296 | 7.38020 | |
| 7 | 04105 | 220.00000 | 3.00000 | 1952.02000 | 2002.86802 | 1017.88226 | 99.85680 | 0.09810 | 5.39363 | 7.57662 | |
| 8 | 04106 | 416.00000 | 1.50000 | 3229.05750 | 3318.46597 | 590.96250 | 60.26881 | 0.10198 | 6.03069 | 8.07995 | |
| Obs | log{AUC | inf} log{C | LF} log{ | LambdaZ} lo | g{Vz_F} Ran | k{Tmax} | Child-E | | | ual Child-P | ugh |
| 1 | 7.1 | 4034 5.06 | 573 | -2.30340 | 7.36913 | 14.0 | | | A | | 5 |
| 2 | 7.4 | 2256 4.78 | 351 | -2.43921 | 7.22272 | 2.0 | | | A | | 5 |
| 3 | 6.9 | 1534 5.29 | 073 | -1.84632 | 7.13705 | 14.0 | | | A | | 5 |
| 4 | 7.6 | 1747 4.58 | 860 | -1.64047 | 6.22907 | 2.0 | | | A | | 6 |
| 5 | 7.7 | 2507 4.48 | 101 | -2.27063 | 6.75163 | 18.0 | | | A | | 5 |
| 6 | 7.3 | 9972 4.80 | 635 | -1.80621 | 6.61256 | 18.0 | | | A | | 5 |
| 7 | 7.6 | 0234 4.60 | 374 | -2.32174 | 6.92548 | 21.5 | | | A | | 5 |
| / | | | | | | | | | | | |
| 4<br>5<br>6 | 7.6<br>7.7<br>7.3 | 1747 4.58<br>2507 4.48<br>9972 4.80 | 860<br>101<br>635 | -1.64047<br>-2.27063<br>-1.80621 | 6.22907<br>6.75163<br>6.61256 | 2.0<br>18.0<br>18.0 | | | A<br>A<br>A | | |

# RAW DATA

### Hepatic Function Group=Moderate

| Obs | Subject<br>ID | Cmax | Tmax | AUCT | AUCinf | Vz_F | Cl_F | LambdaZ | log{Cmax} | log{AUCT} | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 01403 | 207.000 | 00 1.25000 | 960.51333 | 1008.11653 | 1898.74936 | 198.38976 | 0.10448 | 5.33272 | 6.86747 | |
| 10 | 01405 | 259.000 | 00 1.25000 | 1831.00000 | 1870.55382 | 1134.00305 | 106.92021 | 0.09429 | 5.55683 | 7.51262 | |
| 11 | 01407 | 388.000 | 00 1.50000 | 3600.06667 | 3810.94140 | 675.54883 | 52.48047 | 0.07769 | 5.96101 | 8.18871 | |
| 12 | 01409 | 221.000 | 00 1.00000 | 1883.79000 | 2010.53704 | 1368.73641 | 99.47591 | 0.07268 | 5.39816 | 7.54104 | |
| 13 | 04104 | 359.000 | 00 2.00000 | 2689.72500 | 2780.70989 | 806.74296 | 71.92408 | 0.08915 | 5.88332 | 7.89719 | |
| 14 | 04107 | 419.000 | 00 0.75000 | 3096.65500 | 3231.82927 | 774.07373 | 61.88446 | 0.07995 | 6.03787 | 8.03808 | |
| 15 | 04108 | 143.000 | 00 1.75000 | 971.09000 | 986.38429 | 1925.20006 | 202.76073 | 0.10532 | 4.96284 | 6.87842 | |
| 16 | 04110 | 565.000 | 00 1.50000 | 3696.07500 | 3825.60443 | 573.48982 | 52.27932 | 0.09116 | 6.33683 | 8.21503 | |
| Obs | log{AUC | inf} log | {CLF} log{ | LambdaZ} lo | g{Vz_F} Ran | k{Tmax} | Child-F | | Individ | ual Child-P<br>scores | ugh |
| 9 | 6.9 | 1584 5. | 29023 | -2.25872 | 7.54895 | 5.5 | | | В | | 7 |
| 10 | 7.5 | 3399 4. | 67208 | -2.36143 | 7.03351 | 5.5 | | | В | | 8 |
| 11 | 8.2 | 4563 3. | 96044 | -2.55508 | 6.51553 | 8.0 | | | В | | 8 |
| 12 | 7.6 | 0616 4. | 59992 | -2.62173 | 7.22164 | 4.0 | | | В | | 8 |
| 13 | 7.9 | 3046 4. | 27561 | -2.41739 | 6.69301 | 14.0 | | | В | | 7 |
| 14 | 8.0 | 8080 4. | 12527 | -2.52640 | 6.65167 | 2.0 | | | В | | 7 |
| 15 | 6.8 | 9405 5. | 31203 | -2.25076 | 7.56279 | 10.5 | | | В | | 7 |
| 16 | 8.2 | 4947 3. | 95660 | -2.39514 | 6.35174 | 8.0 | | | В | | 7 |

# RAW DATA

### Hepatic Function Group=Healthy

| Obs | Subject<br>ID | Cmax | Tmax | AUCT | AUCinf | Vz_F | Cl_F | LambdaZ | log{Cmax} | log{AUCT} |
|---|---|---|---|---|---|---|---|---|---|---|
| 17 | 00102 | 199.00000 | 4.00000 | 1902.08500 | 1922.96133 | 816.67119 | 104.00625 | 0.12735 | 5.29330 | 7.55071 |
| 18 | 00103 | 307.00000 | 1.75000 | 1863.04750 | 1870.37367 | 703.84229 | 106.93050 | 0.15192 | 5.72685 | 7.52997 |
| 19 | 00104 | 216.00000 | 2.00000 | 1812.21750 | 1831.52555 | 887.40804 | 109.19859 | 0.12305 | 5.37528 | 7.50231 |
| 20 | 00111 | 270.00000 | 2.00000 | 1729.46000 | 1767.45418 | 770.47408 | 113.15711 | 0.14687 | 5.59842 | 7.45556 |
| 21 | 00114 | 189.00000 | 2.50000 | 1112.41750 | 1131.26315 | 1168.42476 | 176.79353 | 0.15131 | 5.24175 | 7.01429 |
| 22 | 00115 | 288.00000 | 2.53333 | 2136.05833 | 2146.74786 | 652.50784 | 93.16418 | 0.14278 | 5.66296 | 7.66672 |
| 23 | 00116 | 149.00000 | 3.00000 | 886.38500 | 916.53880 | 1680.43024 | 218.21226 | 0.12985 | 5.00395 | 6.78715 |
| 24 | 00119 | 192.00000 | 4.00000 | 1706.38150 | 1724.86484 | 957.16011 | 115.95111 | 0.12114 | 5.25750 | 7.44213 |
| Obs | log{AUC | inf} log{( | CLF} log{ | LambdaZ} lo | g{Vz_F} Ranl | k{Tmax} | Child-F | | | ual Child-Pugh<br>scores |
| 17 | 7.5 | 6162 4.64 | 1445 | -2.06079 | 6.70524 | 23.5 | | | | |
| 18 | 7.5 | 3389 4.67 | 7218 | -1.88438 | 6.55655 | 10.5 | | | | |
| 19 | 7.5 | 1290 4.69 | 9317 | -2.09514 | 6.78830 | 14.0 | | | | |
| 20 | 7.4 | 7730 4.72 | 2878 | -1.91823 | 6.64701 | 14.0 | | | | |
| 21 | 7.0 | 3109 5.17 | 7498 | -1.88843 | 7.06341 | 18.0 | | | | |
| 22 | 7.6 | 7171 4.53 | 3436 | -1.94646 | 6.48082 | 20.0 | | | | |
| 23 | 6.8 | 2060 5.38 | 3547 | -2.04134 | 7.42681 | 21.5 | | | | |
| 24 | 7.4 | 5290 4.75 | 317 | -2.11080 | 6.86397 | 23.5 | | | | |

14:27 Thursday, February 8, 2018 4

Algorithme Pharma CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

# DESCRIPTIVE RESULTS (OVERALL)

| Parameter | Hepatic n<br>Function | Min | Mean | Geometric<br>Mean | Median | Max | Range | Standard<br>Deviation | Coefficient |
|---|---|---|---|---|---|---|---|---|---|
| C | Group | 105 0000 | 007 60500 | 061 04455 | 056 50000 | F10 00000 | 202 00000 | 120 52005 | Variation |
| Cmax | Mild 8 | 125.00000 | | | | | | | 46.0774 |
| Cmax | Moderate 8 | 143.00000 | | | | | | | |
| Cmax | Healthy 8 | | | | 207.50000 | | | 55.57942 | 24.5655 |
| Tmax | Mild 8 | 0.75000 | | | | | | 0.82375 | 43.9336 |
| Tmax | Moderate 8 | 0.75000 | | | | | | 0.40089 | |
| Tmax | Healthy 8 | 1.75000 | | | | | | 0.87962 | |
| AUCT | Mild 8 | | 1856.82038 | | | | | | 37.1215 |
| AUCT | Moderate 8 | | 3 2341.11438 | | | | | | 46.6958 |
| AUCT | - | | 1643.50654 | | | | | | 25.7403 |
| AUCinf | | | 9 1899.68370 | | | | | | 37.2124 |
| AUCinf | | | 2440.58459 | | | | | | 47.0102 |
| AUCinf | - | | 1663.96617 | | | | | | 25.1680 |
| Vz_F | Mild 8 | | 991.26784 | | | | | 386.04048 | 38.9441 |
| Vz_F | Moderate 8 | | 2 1144.56803 | | | | | 537.99098 | 47.0038 |
| Vz_F | Healthy 8 | | | | | | 1027.92241 | | 35.0606 |
| CL_F | Mild 8 | 60.26883 | 118.19988 | 111.58768 | 109.68998 | 198.48916 | 138.22035 | 43.20623 | 36.5535 |
| CL_F | Moderate 8 | 52.27932 | 105.76437 | 92.20576 | 85.69999 | 202.76073 | 150.48141 | 61.87438 | 58.5021 |
| CL_F | Healthy 8 | 93.16418 | 3 129.67669 | 124.37731 | 111.17785 | 218.21226 | 125.04808 | 43.83200 | 33.8010 |
| LambdaZ | Mild 8 | 0.08723 | 0.12581 | 0.12077 | 0.10262 | 0.19389 | 0.10666 | 0.03990 | 31.7121 |
| LambdaZ | Moderate 8 | 0.07268 | 0.08934 | 0.08863 | 0.09016 | 0.10532 | 0.03264 | 0.01204 | 13.4733 |
| LambdaZ | Healthy 8 | 0.12114 | 0.13679 | 0.13626 | 0.13632 | 0.15192 | 0.03078 | 0.01281 | 9.3622 |
| 1Cmax | Mild 8 | 4.8283 | L 5.56546 | | 5.54711 | 6.24998 | 1.42166 | 0.47671 | 8.5655 |
| 1Cmax | Moderate 8 | 4.96284 | 5.68370 | | 5.72008 | 6.33683 | 1.37398 | 0.44868 | 7.8942 |
| 1Cmax | Healthy 8 | 5.0039 | 5.39500 | | 5.33429 | 5.72685 | 0.72290 | 0.24766 | 4.5906 |
| lauct | Mild 8 | 6.8860 | 7.46821 | | 7.48636 | 8.07995 | 1.19387 | 0.36606 | 4.9016 |
| lauct | Moderate 8 | 6.8674 | 7.64232 | | 7.71912 | 8.21503 | 1.34756 | 0.54237 | 7.0969 |
| lauct | Healthy 8 | 6.7871 | 7.36860 | | 7.47894 | 7.66672 | 0.87957 | 0.30297 | 4.1117 |
| lAUCinf | Mild 8 | 6.91534 | 7.49126 | | 7.51245 | 8.10726 | 1.19192 | 0.36456 | 4.8664 |
| lAUCinf | Moderate 8 | 6.8940 | 7.68205 | | 7.76831 | 8.24947 | 1.35543 | 0.54720 | 7.1231 |
| lAUCinf | Healthy 8 | 6.82060 | 7.38275 | | 7.49510 | 7.67171 | 0.85110 | 0.29491 | 3.9946 |
| lCLF | Mild 8 | 4.09883 | L 4.71481 | | 4.69362 | 5.29073 | 1.19192 | 0.36456 | 7.7322 |
| 1CLF | Moderate 8 | 3.95660 | 4.52402 | | 4.43776 | 5.31203 | 1.35543 | 0.54720 | 12.0955 |
| 1CLF | Healthy 8 | 4.53436 | 4.82332 | | 4.71097 | 5.38547 | 0.85110 | 0.29491 | 6.1143 |
| lLambdaZ | Mild 8 | -2.43921 | -2.11386 | | -2.27678 | -1.64047 | 0.79874 | 0.29964 | -14.1749 |
| lLambdaZ | Moderate 8 | -2.62173 | -2.42333 | | -2.40627 | -2.25076 | 0.37097 | 0.13569 | -5.5994 |
| lLambdaZ | Healthy 8 | -2.11080 | -1.99319 | | -1.99390 | -1.88438 | 0.22643 | 0.09391 | -4.7114 |
| lVz F | Mild 8 | 6.2290 | | | 6.83856 | | | 0.40774 | 5.9709 |
| lVz F | Moderate 8 | 6.35174 | | | 6.86326 | | | 0.46548 | |
| lVz F | Healthy 8 | 6.48082 | | | 6.74677 | | | 0.30656 | |
| RkTmax | Mild 8 | 2.00000 | | | | | | 7.42552 | |
| RkTmax | Moderate 8 | 2.00000 | | | | | | 3.80730 | |
| RkTmax | Healthy 8 | 10.50000 | | | | 23.50000 | | 4.85320 | 26.7763 |
| MINITIMA | incurcing 0 | 10.50000 | , 10.12300 | 17.50005 | 17.00000 | 23.30000 | 13.00000 | 4.05520 | 20.7703 |

## ----- SUMMARY REPORT -----

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

#### ANOVA analysis

----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=1 Param=Cmax

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components
Group Effect FunctionGroup
Estimation Method REML

Residual Variance Method None

Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 3 1 2 3

#### Dimensions

Covariance Parameters Columns in X 4 Columns in Z Subjects 0 24 Max Obs per Subject

#### Number of Observations

Number of Observations Read 24 Number of Observations Used 24 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 265.15407978 1 259.49486652 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup 1 17564 Residual FunctionGroup 2 19084 Residual FunctionGroup 3 3089.07

#### Fit Statistics

-2 Res Log Likelihood 259.5 AIC (Smaller is Better) 265.5 AICC (Smaller is Better) 266.9 BIC (Smaller is Better) 269.0

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 2 5.66 0.0590

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F DF DF

FunctionGroup 2 21 2.05 0.1536

----- SUMMARY REPORT -----Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis

----- SUMMARY REPORT -----

The Mixed Procedure

Order=1 Param=Cmax

Least Squares Means

Effect Hepatic Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error Group 287.62 46.856521 6.14 <.0001 0.1207.00368.25 FunctionGroup 1 320.13 48.842121 6.55 <.0001 0.1236.08404.17 FunctionGroup 2 FunctionGroup 3 226.25 19.6503 21 11.51 <.0001 0.1 192.44 260.06

Differences of Least Squares Means

Effect Hepatic Hepatic Estimate Standard DF t Value Pr > |t| Adjustment Adj P Alpha Lower Upper Function Function Error Group Group -32.5000 67.683721 -0.48 0.6361 Tukey-Kramer 0.8814 0.1 -148.9783.9663 FunctionGroup 1 2 3 61.3750 50.8101 21 1.21 0.2405 Tukey-Kramer 0.4617 0.1 -26.0561 148.81 FunctionGroup 1 3 93.8750 52.6468 21 1.78 0.0890 Tukey-Kramer 0.1995 0.1 3.2834 184.47 FunctionGroup 2

> Differences of Least Squares Means Hepatic Hepatic Adj Effect Adi Function Function Lower Upper Group Group FunctionGroup 1 2 -179.37 114.37 FunctionGroup 1 3 -48.8797 171.63 FunctionGroup 2 3 -20.3652 208.12

## ----- SUMMARY REPORT -----

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

#### ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=3 Param=AUCT

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Estimation Method REML

Residual Variance Method None

Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 3 1 2 3

#### Dimensions

Covariance Parameters Columns in X 4 Columns in Z Subjects 0 24 Max Obs per Subject

#### Number of Observations

Number of Observations Read 24 Number of Observations Used 24 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 345.79800104

1 1 339.95357919 0.00000000

#### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup 1 475106 Residual FunctionGroup 2 1195091 Residual FunctionGroup 3 178966

#### Fit Statistics

-2 Res Log Likelihood 340.0 AIC (Smaller is Better) 346.0 AICC (Smaller is Better) 347.4 BIC (Smaller is Better) 349.5

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 2 5.84 0.0538

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F DF DF

FunctionGroup 2 21 1.51 0.2436

----- SUMMARY REPORT -----Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis

----- SUMMARY REPORT -----

The Mixed Procedure

Order=3 Param=AUCT

Least Squares Means

Effect Hepatic Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error Group FunctionGroup 1 1856.82 243.70 21 7.62 <.0001 0.1 1437.48 2276.16 2341.11 386.5121 6.06 <.0001 0.11676.043006.19 FunctionGroup 2 FunctionGroup 3 1643.51 149.57 21 10.99 <.0001 0.1 1386.14 1900.88

Differences of Least Squares Means

Effect Hepatic Hepatic Estimate Standard DF t Value Pr > |t| Adjustment Adj P Alpha Lower Upper Function Function Error Group Group -484.29 456.92 21 -1.06 0.3012 Tukey-Kramer 0.5486 0.1 -1270.53 301.95 FunctionGroup 1 2 3 213.31 285.94 21 0.75 0.4639 Tukey-Kramer 0.7393 0.1 -278.71 705.33 FunctionGroup 1 697.61 414.44 21 1.68 0.1071 Tukey-Kramer 0.2348 0.1 -15.5299 1410.75 3 FunctionGroup 2

> Differences of Least Squares Means Hepatic Hepatic Adj Effect Adj Function Function Lower Upper Group Group FunctionGroup 1 2 -1475.78 507.19 FunctionGroup 1 3 -407.15 833.77 FunctionGroup 2 3 -201.69 1596.91

## ----- SUMMARY REPORT -----

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

#### ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=4 Param=AUCinf

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components
Group Effect FunctionGroup
Estimation Method REML

Residual Variance Method None

Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 3 1 2 3

#### Dimensions

Covariance Parameters Columns in X 4 Columns in Z Subjects 0 24 Max Obs per Subject

#### Number of Observations

Number of Observations Read 24 Number of Observations Used 24 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 347.35488834

1 1 340.84221814 0.00000000

#### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup 1 499733 Residual FunctionGroup 2 1316350 Residual FunctionGroup 3 175382

#### Fit Statistics

-2 Res Log Likelihood 340.8 AIC (Smaller is Better) 346.8 AICC (Smaller is Better) 348.3 BIC (Smaller is Better) 350.4

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 2 6.51 0.0385

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F DF DF

FunctionGroup 2 21 1.74 0.1991

14:27 Thursday, February 8, 2018 10

Algorithme Pharma

53: Effect of Menatic Tennil CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis

----- SUMMARY REPORT -----

The Mixed Procedure

Order=4 Param=AUCinf

Least Squares Means

| Effect | Function | | Standard DF t<br>Error | Value P | r > t A | lpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| | Group | | | | | | | |
| FunctionGroup | 1 | 1899.68 | 249.93 21 | 7.60 | <.0001 | 0.11 | 469.61 | 2329.75 |
| FunctionGroup | 2 | 2440.58 | 405.64 21 | 6.02 | <.0001 | 0.11 | 742.58 | 3138.59 |
| FunctionGroup | 3 | 1663.97 | 148.06 21 | 11.24 | < .0001 | 0.11 | 409.19 | 1918.75 |

### Differences of Least Squares Means

| Effect | Hepatic | Hepatic | Estimate | Standard DF t | Value Pr | > t | Adjustment | Adj I | P Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Function | Function | | Error | | | | | | | |
| | Group | Group | | | | | | | | | |
| FunctionGroup | 1 | 2 | -540.90 | 476.46 21 | -1.14 | 0.2691 | Tukey-Kramer | 0.5037 | 7 0.1 | -1360.76 | 278.96 |
| FunctionGroup | 1 | 3 | 235.72 | 290.50 21 | 0.81 | 0.4262 | Tukey-Kramer | 0.7002 | 2 0.1 | -264.16 | 735.59 |
| FunctionGroup | 2 | 3 | 776.62 | 431.82 21 | 1.80 | 0.0865 | Tukev-Kramer | 0.1944 | 4 0.1 | 33.5712 | 1519.67 |

| Differer | nces of Le | east Squa | res Means | |
|---------------|------------|-----------|-----------|---------|
| Effect | Hepatic | Hepatic | Adj | Adj |
| | Function | Function | Lower | Upper |
| | Group | Group | | |
| FunctionGroup | 1 | 2 | -1574.78 | 492.98 |
| FunctionGroup | 1 | 3 | -394.65 | 866.08 |
| FunctionGroup | 2 | 3 | -160.40 | 1713.64 |

#### ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=8 Param=1Cmax

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Dependent Variable Value
Covariance Structure Variance Components
Group Effect FunctionGroup
Estimation Method REML

Residual Variance Method None

Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 3 1 2 3

#### Dimensions

Covariance Parameters 3 Columns in X 4 Columns in Z Subjects 0 24 Max Obs per Subject

#### Number of Observations

Number of Observations Read 24 Number of Observations Used 24 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 27.77835282

1 1 24.70196938 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup 1 0.2273 Residual FunctionGroup 2 0.2013 Residual FunctionGroup 3 0.06134

#### Fit Statistics

-2 Res Log Likelihood 24.7 AIC (Smaller is Better) 30.7 AICC (Smaller is Better) 32.1 BIC (Smaller is Better) 34.2

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 2 3.08 0.2148

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F DF DF

FunctionGroup 2 21 1.42 0.2630

14:27 Thursday, February 8, 2018 12

Algorithme Pharma

153: Effect of Henatic Transformers CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis

----- SUMMARY REPORT -----

The Mixed Procedure

Order=8 Param=1Cmax

Least Squares Means

| | | шса. | oc bquareb me | aiib | | |
|---|---|---|---|---|---|---|
| Effect | Hepatic<br>Function<br>Group | | Standard DF t<br>Error | Value P | r > t A | lpha Lower Upper |
| FunctionGroup | 1 | 5.5655 | 0.1685 21 | 33.02 | <.0001 | 0.15.27545.8555 |
| FunctionGroup | 2 | 5.6837 | 0.1586 21 | 35.83 | < .0001 | 0.15.41075.9567 |
| FunctionGroup | 3 | 5.3950 | 0.08756 21 | 61.61 | < .0001 | 0.15.24435.5457 |

### Differences of Least Squares Means

| Effect | Hepatic | Hepatic | Estimate | Standard DF | t Value Pr | > t | Adjustment | Adj I | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Function | Function | | Error | | | | | | | |
| | Group | Group | | | | | | | | | |
| FunctionGroup | 1 | 2 | -0.1182 | 0.2315 21 | -0.51 | 0.6148 | Tukey-Kramer | 0.8669 | 0.1 | -0.5165 | 0.2800 |
| FunctionGroup | 1 | 3 | 0.1705 | 0.1899 21 | 0.90 | 0.3796 | Tukey-Kramer | 0.6478 | 0.1 | -0.1564 | 0.4973 |
| FunctionGroup | 2 | 3 | 0.2887 | 0.1812 21 | 1.59 | 0.1260 | Tukev-Kramer | 0.2704 | 1 0.1 | -0.02309 | 0.6005 |

| Differenc | es | of | Lea | ast | Squares | Means | |
|-----------|-----|-----|-----|-----|---------|-------|-----|
| Effect | Her | at. | ic | Her | patic | Adi | Adi |

| Ellect | перастс | перастс | Auj | Adj |
|---------------|----------|----------|---------|--------|
| | Function | Function | Lower | Upper |
| | Group | Group | | |
| FunctionGroup | 1 | 2 | -0.6205 | 0.3840 |
| FunctionGroup | 1 | 3 | -0.2417 | 0.5826 |
| FunctionGroup | 2 | 3 | -0.1045 | 0.6819 |

#### ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=9 Param=1AUCT

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components
Group Effect FunctionGroup
Estimation Method REML

Residual Variance Method None

Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 3 1 2 3

#### Dimensions

Covariance Parameters 3 Columns in X 4 Columns in Z Subjects 0 24 Max Obs per Subject

#### Number of Observations

Number of Observations Read 24 Number of Observations Used 24 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 29.02854090

1 1 26.48128492 0.00000000

#### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup 1 0.1340 Residual FunctionGroup 2 0.2942 Residual FunctionGroup 3 0.09179

#### Fit Statistics

-2 Res Log Likelihood 26.5 AIC (Smaller is Better) 32.5 AICC (Smaller is Better) 33.9 BIC (Smaller is Better) 36.0

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 2 2.55 0.2798

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F DF DF

FunctionGroup 2 21 0.80 0.4626

14:27 Thursday, February 8, 2018 14

Algorithme Pharma CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis

----- SUMMARY REPORT -----

The Mixed Procedure

Order=9 Param=1AUCT

Least Squares Means

| nease squares means | | | | | | |
|---|---|---|---|---|---|---|
| Effect | Hepatic<br>Function<br>Group | | tandard DF t<br>Error | Value P | r > t A | lpha Lower Upper |
| FunctionGroup | 1 | 7.4682 | 0.1294 21 | 57.70 | < .0001 | 0.17.24557.6909 |
| FunctionGroup | 2 | 7.6423 | 0.1918 21 | 39.85 | < .0001 | 0.17.31247.9723 |
| FunctionGroup | 3 | 7.3686 | 0.1071 21 | 68.79 | < .0001 | 0.17.18437.5529 |

### Differences of Least Squares Means

| Effect | Hepatic | Hepatic | Estimate S | tandard DF t | Value Pr | : > t | Adjustment | Adj PAl | lpha Lowe | er Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| | Function | Function | | Error | | | | | | |
| | Group | Group | | | | | | | | |
| FunctionGroup | 1 | 2 | -0.1741 | 0.2313 21 | -0.75 | 0.4600 | Tukey-Kramer | 0.7354 | 0.1 -0.572 | 22 0.2240 |
| FunctionGroup | 1 | 3 | 0.09961 | 0.1680 21 | 0.59 | 0.5596 | Tukey-Kramer | 0.8254 | 0.1 -0.189 | 95 0.3887 |
| FunctionGroup | 2 | 3 | 0.2737 | 0.2196 21 | 1.25 | 0.2264 | Tukev-Kramer | 0.4402 | 0.1-0.104 | 2 0.6517 |

| Differenc | es of Lea | ast Square | es Means | |
|---------------|-----------|------------|----------|--------|
| Effect | Hepatic | Hepatic | Adj | Adj |
| | Function | Function | Lower | Upper |
| | Group | Group | | |
| FunctionGroup | 1 | 2 | -0.6761 | 0.3279 |
| FunctionGroup | 1 | 3 | -0.2649 | 0.4642 |
| FunctionGroup | 2 | 3 | -0.2029 | 0.7503 |

#### CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

#### ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=10 Param=lAUCinf

#### Model Information

Data Set WORK.KINDATA

Value Dependent Variable

Covariance Structure Variance Components
Group Effect FunctionGroup
Estimation Method REML

Residual Variance Method None

Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 3 1 2 3

#### Dimensions

Covariance Parameters 3 Columns in X 4 Columns in Z Subjects 0 24 Max Obs per Subject

#### Number of Observations

Number of Observations Read 24 Number of Observations Used Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 29.00237589

1 1 26.17053116 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup 1 0.1329 Residual FunctionGroup 2 0.2994 Residual FunctionGroup 3 0.08697

#### Fit Statistics

-2 Res Log Likelihood 26.2 AIC (Smaller is Better) 32.2 AICC (Smaller is Better) 33.6 BIC (Smaller is Better) 35.7

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 2 2.83 0.2427

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F DF DF

FunctionGroup 2 21 0.96 0.3987

14:27 Thursday, February 8, 2018 16

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis

----- SUMMARY REPORT -----

#### The Mixed Procedure

### Order=10 Param=lAUCinf

#### Least Squares Means

| Effect | Hepatic | Estimate | Standard DF t | Value 1 | Pr > t | Alpha Lower | Upper |
|---|---|---|---|---|---|---|---|
| | Function | | Error | | | | |
| | Group | | | | | | |
| FunctionGroup | 1 | 7.4913 | 0.1289 21 | 58.12 | <.0001 | 0.17.2695 | 7.7130 |
| FunctionGroup | 2 | 7.6821 | 0.1935 21 | 39.71 | <.0001 | 0.17.3491 | 8.0150 |
| FunctionGroup | 3 | 7.3828 | 0.1043 21 | 70.81 | <.0001 | 0.17.2033 | 7.5622 |

### Differences of Least Squares Means

| Effect | Hepatic | Hepatic | Estimate | Standard DF | t Value Pr | > t | Adjustment | Adj P | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Function | Function | | Error | | | | | | | |
| | Group | Group | | | | | | | | | |
| FunctionGroup | 1 | 2 | -0.1908 | 0.2325 21 | -0.82 | 0.4210 | Tukey-Kramer | 0.6946 | 0.1 | -0.5908 | 0.2092 |
| FunctionGroup | 1 | 3 | 0.1085 | 0.1658 21 | 0.65 | 0.5199 | Tukey-Kramer | 0.7919 | 0.1 | -0.1768 | 0.3938 |
| FunctionGroup | 2 | 3 | 0.2993 | 0.2198 21 | 1.36 | 0.1877 | Tukev-Kramer | 0.3783 | 0.1 | -0.07888 ( | 0.6775 |

| Differences of Least Squares M | s Means |
|--------------------------------|---------|
|--------------------------------|---------|

| Effect | Hepatic | Hepatic | Adj | Adj |
|---------------|----------|----------|---------|--------|
| | Function | Function | Lower | Upper |
| | Group | Group | | |
| FunctionGroup | 1 | 2 | -0.6952 | 0.3137 |
| FunctionGroup | 1 | 3 | -0.2512 | 0.4683 |
| FunctionGroup | 2 | 3 | -0.1776 | 0.7762 |

14:27 Thursday, February 8, 2018 17

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis Geometric LSmeans -----SUMMARY REPORT -----

| Obs | Parameters | Group | GeoLSmeans |
|-----|------------|----------|------------|
| 1 | 1Cmax | Mild | 261.24 |
| 2 | 1Cmax | Moderate | 294.03 |
| 3 | 1Cmax | Normal | 220.30 |
| 4 | lauct | Mild | 1751.47 |
| 5 | lauct | Moderate | 2084.57 |
| 6 | lauct | Normal | 1585.42 |
| 7 | lAUCinf | Mild | 1792.31 |
| 8 | lAUCinf | Moderate | 2169.06 |
| 9 | lAUCinf | Normal | 1608.01 |

14:27 Thursday, February 8, 2018 18

Algorithme Pharma

Signature 13:28 Thursday, February 8, 2018 18

Algorithme Pharma CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

ANOVA analysis
RATIO ESTIMATE BASED ON ln-TRANSFORMED PARAMETERS
----- SUMMARY REPORT -----

| Obs | Parameters | Group vs | | Adj<br>P-value | | L90 | U90 |
|---|---|---|---|---|---|---|---|
| 1 | 1Cmax | 1 | 2 | 0.8669 | 88.848 | 53.769 | 146.815 |
| 2 | 1Cmax | 1 | 3 | 0.6478 | 118.585 | 78.531 | 179.068 |
| 3 | 1Cmax | 2 | 3 | 0.2704 | 133.469 | 90.079 | 197.759 |
| 4 | lauct | 1 | 2 | 0.7354 | 84.021 | 50.859 | 138.804 |
| 5 | lauct | 1 | 3 | 0.8254 | 110.474 | 76.725 | 159.067 |
| 6 | lAUCT | 2 | 3 | 0.4402 | 131.484 | 81.636 | 211.770 |
| 7 | lAUCinf | 1 | 2 | 0.6946 | 82.631 | 49.896 | 136.842 |
| 8 | lAUCinf | 1 | 3 | 0.7919 | 111.462 | 77.784 | 159.720 |
| 9 | lAUCinf | 2 | 3 | 0.3783 | 134.891 | 83.728 | 217.318 |

## ----- SUMMARY REPORT -----

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=AUCT

Number of Observations Read Number of Observations Used Number of Observations with Missing Values  $\,$  8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

1 1007220 1007220 1.21 0.2893 Model

14 11622321 830166 Error

Corrected Total 15 12629542

Root MSE 911.13435 R-Square 0.0798 Dependent Mean 2098.96738 Adj R-Sq 0.0140 Coeff Var 43.40870

#### Parameter Estimates

Variable DF Parameter Standard t Value Pr > |t| 95% Confidence Limits Estimate Error

Intercept 1 791.05592 1209.05488 0.65 0.5235 -1802.10890 3384.22073 indiv 1 209.26583 189.98465 1.10 0.2893 -198.21071 616.74237 CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

### NAME OF FORMER VARIABLE=AUCT

#### Output Statistics

| | | | - | out Statis | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent | | | Residual | Std Error | | -2-1 | 0 1 2 | Cook's |
| | Variable | | Mean Predict | | Residual | Residual | | | D |
| 1 | 1229 | 1837 | 329.0631 | -608.0676 | 849.6 | -0.716 | * | | 0.038 |
| 2 | 1630 | 1837 | 329.0631 | -207.7826 | 849.6 | -0.245 | | | 0.004 |
| 3 | 978.5525 | 1837 | 329.0631 | -858.8326 | 849.6 | -1.011 | ** | | 0.077 |
| 4 | 2020 | 2047 | 232.6827 | -26.8759 | 880.9 | -0.0305 | | | 0.000 |
| 5 | 2212 | 1837 | 329.0631 | 374.9404 | 849.6 | 0.441 | | | 0.015 |
| 6 | 1604 | 1837 | 329.0631 | -233.4726 | 849.6 | -0.275 | | | 0.006 |
| 7 | 1952 | 1837 | 329.0631 | 114.6349 | 849.6 | 0.135 | | | 0.001 |
| 8 | 3229 | 1837 | 329.0631 | 1392 | 849.6 | 1.638 | 1 | *** | 0.201 |
| 9 | 960.5133 | 2256 | 268.6789 | -1295 | 870.6 | -1.488 | ** | | 0.105 |
| 10 | 1831 | 2465 | 403.0183 | -634.1826 | 817.2 | -0.776 | * | | 0.073 |
| 11 | 3600 | 2465 | 403.0183 | 1135 | 817.2 | 1.389 | | ** | 0.235 |
| 12 | 1884 | 2465 | 403.0183 | -581.3926 | 817.2 | -0.711 | * | | 0.062 |
| 13 | 2690 | 2256 | 268.6789 | 433.8082 | 870.6 | 0.498 | | | 0.012 |
| 14 | 3097 | 2256 | 268.6789 | 840.7382 | 870.6 | 0.966 | | * | 0.044 |
| 15 | 971.0900 | 2256 | 268.6789 | -1285 | 870.6 | -1.476 | ** | | 0.104 |
| 16 | 3696 | 2256 | 268.6789 | 1440 | 870.6 | 1.654 | | *** | 0.130 |
| 17 | 1902 | | | | | | | | |
| 18 | 1863 | | | | | | | | |
| 19 | 1812 | | | | | | | | |
| 20 | 1729 | | | | | | | | |
| 21 | 1112 | | | | | | | | |
| 22 | 2136 | | | | | | | | |
| 23 | 886.3850 | | | | | | | | |
| 23 | 1706 | | | | | | | | |
| 24 | 1706 | | | | | | | | |

Sum of Residuals 0 Sum of Squared Residuals 11622321 Predicted Residual SS (PRESS) 15048631 Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=AUCinf

Number of Observations Read Number of Observations Used Number of Observations with Missing Values  $\,$  8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

1 1254768 1254768 1.39 0.2579 Model

14 12628107 902008 Error

Corrected Total 15 13882875

Root MSE 949.74084 R-Square 0.0904 Dependent Mean 2170.13414 Adj R-Sq 0.0254 Coeff Var 43.76415

#### Parameter Estimates

Variable DF Parameter Standard t Value Pr > |t| 95% Confidence Limits

Estimate Error

Intercept 1 710.31943 1260.28482 0.56 0.5819 -1992.72268 3413.36153 indiv 1 233.57035 198.03465 1.18 0.2579 -191.17173 658.31244

### CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=AUCinf

### Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 1262 | 1878 | 343.0061 | -616.3133 | 885.6 | -0.696 | * | | 0.036 |
| 2 | 1673 | 1878 | 343.0061 | -204.8552 | 885.6 | -0.231 | | | 0.004 |
| 3 | 1008 | 1878 | 343.0061 | -870.5595 | 885.6 | -0.983 | * | | 0.072 |
| 4 | 2033 | 2112 | 242.5419 | -78.3261 | 918.2 | -0.0853 | | | 0.000 |
| 5 | 2264 | 1878 | 343.0061 | 386.2334 | 885.6 | 0.436 | | | 0.014 |
| 6 | 1636 | 1878 | 343.0061 | -242.6412 | 885.6 | -0.274 | | | 0.006 |
| 7 | 2003 | 1878 | 343.0061 | 124.6968 | 885.6 | 0.141 | | | 0.001 |
| 8 | 3318 | 1878 | 343.0061 | 1440 | 885.6 | 1.626 | | *** | 0.198 |
| 9 | 1008 | 2345 | 280.0633 | -1337 | 907.5 | -1.473 | ** | | 0.103 |
| 10 | 1871 | 2579 | 420.0949 | -708.3284 | 851.8 | -0.832 | * | | 0.084 |
| 11 | 3811 | 2579 | 420.0949 | 1232 | 851.8 | 1.446 | | ** | 0.254 |
| 12 | 2011 | 2579 | 420.0949 | -568.3452 | 851.8 | -0.667 | * | | 0.054 |
| 13 | 2781 | 2345 | 280.0633 | 435.3980 | 907.5 | 0.480 | | | 0.011 |
| 14 | 3232 | 2345 | 280.0633 | 886.5174 | 907.5 | 0.977 | | * | 0.045 |
| 15 | 986.3843 | 2345 | 280.0633 | -1359 | 907.5 | -1.497 | ** | | 0.107 |
| 16 | 3826 | 2345 | 280.0633 | 1480 | 907.5 | 1.631 | | *** | 0.127 |
| 17 | 1923 | | | | | | | | |
| 18 | 1870 | | | | | | | | |
| 19 | 1832 | | | | | | | | |
| 20 | 1767 | | | | | | | | |
| 21 | 1131 | | | | | | | | |
| 22 | 2147 | | | | | | | | |
| 23 | 916.5388 | | | | | | | | |
| 24 | 1725 | | | | | | | | |

Sum of Residuals Sum of Squared Residuals 12628107 Predicted Residual SS (PRESS) 16386093 Algorithme Pharma

#### CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=CL F

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source Model 1572.52895 1572.52895 0.57 0.4644

Error 14 38913 2779.46872

Corrected Total 15 40485

Root MSE 52.72067 R-Square 0.0388 Dependent Mean 111.98212 Adj R-Sq -0.0298 Coeff Var 47.07954

Parameter Estimates

 Variable
 DF Parameter Standard t Estimates
 Value Pr > |t|
 95% Confidence Limits

 Intercept
 1 163.66128 69.95914
 2.34 0.0347
 13.61384 313.70872

 indiv
 1 -8.26867 10.99302
 -0.75 0.4644 -31.84635
 15.30902

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=CL F

### Output Statistics

| D | D 32 3 | _ | | | Q+ | 0 1 | 0 1 0 | G = -1-1 = |
|---|---|---|---|---|---|---|---|---|
| _ | | | | | | -2-1 | . 0 1 2 | Cook's<br>D |
| 158.4964 | 122.3180 | 19.0405 | 36.1785 | 49.162 | 0.736 | 1 | * | 0.041 |
| 119.5232 | 122.3180 | 19.0405 | -2.7948 | 49.162 | -0.0568 | | | 0.000 |
| 198.4892 | 122.3180 | 19.0405 | 76.1712 | 49.162 | 1.549 | | *** | 0.180 |
| 98.3567 | 114.0493 | 13.4636 | -15.6926 | 50.973 | -0.308 | | | 0.003 |
| 88.3234 | 122.3180 | 19.0405 | -33.9945 | 49.162 | -0.691 | * | | 0.036 |
| 122.2845 | 122.3180 | 19.0405 | -0.0334 | 49.162 | -0.0007 | | | 0.000 |
| 99.8568 | 122.3180 | 19.0405 | -22.4611 | 49.162 | -0.457 | | | 0.016 |
| 60.2688 | 122.3180 | 19.0405 | -62.0491 | 49.162 | -1.262 | ** | | 0.119 |
| 198.3898 | 105.7806 | 15.5465 | 92.6091 | 50.376 | 1.838 | | *** | 0.161 |
| 106.9202 | 97.5120 | 23.3197 | 9.4082 | 47.283 | 0.199 | | | 0.005 |
| 52.4805 | 97.5120 | 23.3197 | -45.0315 | 47.283 | -0.952 | * | | 0.110 |
| 99.4759 | 97.5120 | 23.3197 | 1.9640 | 47.283 | 0.0415 | | | 0.000 |
| 71.9241 | 105.7806 | 15.5465 | -33.8565 | 50.376 | -0.672 | * | | 0.022 |
| 61.8845 | 105.7806 | 15.5465 | -43.8962 | 50.376 | -0.871 | * | | 0.036 |
| 202.7607 | 105.7806 | 15.5465 | 96.9801 | 50.376 | 1.925 | | *** | 0.176 |
| 52.2793 | 105.7806 | 15.5465 | -53.5013 | 50.376 | -1.062 | ** | | 0.054 |
| 104.0063 | | | | | | | | |
| 106.9305 | | | | | | | | |
| 109.1986 | | | | | | | | |
| 113.1571 | | | | | | | | |
| 176.7935 | | | | | | | | |
| 93.1642 | | | | | | | | |
| 218.2123 | | | | | | | | |
| 115.9511 | | | | | | | | |
| | Variable 158.4964 119.5232 198.4892 98.3567 88.3234 122.2845 99.8568 60.2688 198.3898 106.9202 52.4805 99.4759 71.9241 61.8845 202.7607 52.2793 104.0063 106.9305 109.1986 113.1571 176.7935 93.1642 218.2123 | Variable Value 158.4964 122.3180 119.5232 122.3180 98.3567 114.0493 88.3234 122.3180 122.2845 122.3180 99.8568 122.3180 60.2688 122.3180 198.3898 105.7806 106.9202 97.5120 99.4759 97.5120 71.9241 105.7806 61.8845 105.7806 202.7607 105.7806 52.2793 105.7806 104.0063 106.9305 109.1986 113.1571 176.7935 93.1642 218.2123 | Dependent Variable Value Std Error Mean Variable Value Mean Predict 158.4964 122.3180 19.0405 119.5232 122.3180 19.0405 198.4892 122.3180 19.0405 98.3567 114.0493 13.4636 88.3234 122.3180 19.0405 122.2845 122.3180 19.0405 99.8568 122.3180 19.0405 60.2688 122.3180 19.0405 198.3898 105.7806 15.5465 106.9202 97.5120 23.3197 99.4759 97.5120 23.3197 71.9241 105.7806 15.5465 202.7607 105.7806 15.5465 52.2793 105.7806 15.5465 104.0063 106.9305 109.1986 113.1571 176.7935 93.1642 218.2123 188.2123 | Dependent Predicted Value Mean Predict 158.4964 122.3180 19.0405 36.1785 119.5232 122.3180 19.0405 76.1712 98.3567 114.0493 13.4636 -15.6926 88.3234 122.3180 19.0405 -33.9945 122.2845 122.3180 19.0405 -0.0334 99.8568 122.3180 19.0405 -0.0334 99.8568 122.3180 19.0405 -22.4611 60.2688 122.3180 19.0405 -62.0491 198.3898 105.7806 15.5465 92.6091 106.9202 97.5120 23.3197 9.4082 52.4805 97.5120 23.3197 -45.0315 99.4759 97.5120 23.3197 1.9640 71.9241 105.7806 15.5465 -33.8565 61.8845 105.7806 15.5465 -43.8962 202.7607 105.7806 15.5465 -53.5013 104.0063 106.9305 109.1986 113.1571 176.7935 93.1642 218.2123 | Dependent Predicted Value Mean Predict Residual Std Error Residual 158.4964 122.3180 19.0405 36.1785 49.162 119.5232 122.3180 19.0405 -2.7948 49.162 198.4892 122.3180 19.0405 76.1712 49.162 98.3567 114.0493 13.4636 -15.6926 50.973 88.3234 122.3180 19.0405 -33.9945 49.162 122.2845 122.3180 19.0405 -0.0334 49.162 99.8568 122.3180 19.0405 -0.0334 49.162 99.8568 122.3180 19.0405 -22.4611 49.162 198.3898 105.7806 15.5465 92.6091 50.376 106.9202 97.5120 23.3197 9.4082 47.283 52.4805 97.5120 23.3197 9.4082 47.283 99.4759 97.5120 23.3197 1.9640 47.283 71.9241 105.7806 15.5465 -33.8565 50.376 61.8845 105.7806 15.5465 -33.8565 50.376 61.8845 105.7806 15.5465 -33.8565 50.376 202.7607 105.7806 15.5465 -53.5013 50.376 104.0063 106.9305 109.1986 113.1571 176.7935 93.1642 218.2123 | Dependent Variable Value Mean Error Predict Residual Residual Student Residual 158.4964 122.3180 19.0405 36.1785 49.162 0.736 119.5232 122.3180 19.0405 -2.7948 49.162 -0.0568 198.4892 122.3180 19.0405 76.1712 49.162 1.549 98.3567 114.0493 13.4636 -15.6926 50.973 -0.308 88.3234 122.3180 19.0405 -33.9945 49.162 -0.691 122.2845 122.3180 19.0405 -0.0334 49.162 -0.0007 99.8568 122.3180 19.0405 -22.4611 49.162 -0.457 60.2688 122.3180 19.0405 -62.0491 49.162 -0.457 60.2688 122.3180 19.0405 -62.0491 49.162 -0.457 60.2688 122.3180 19.0405 -62.0491 49.162 -0.457 198.3898 105.7806 15.5465 92.6091 50.376 1.838 </td <td> Dependent Predicted Std Error Residual Std Error Student Residual Residual Residual Std Error Student Residual Residual Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Student Std Error Stdent Std Error Student Std Error Stdent Std Error Student Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Std Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Error Stdent Std Erro</td> <td>Variable Value Mean Predict Residual Residual 158.4964 122.3180 19.0405 36.1785 49.162 0.736 * 119.5232 122.3180 19.0405 -2.7948 49.162 -0.0568 198.4892 122.3180 19.0405 76.1712 49.162 1.549 *** 98.3567 114.0493 13.4636 -15.6926 50.973 -0.308 *** 88.3234 122.3180 19.0405 -33.9945 49.162 -0.691 * ** 122.2845 122.3180 19.0405 -0.0334 49.162 -0.457 ** 60.2688 122.3180 19.0405 -22.4611 49.162 -0.457 ** 60.2688 122.3180 19.0405 -62.0491 49.162 -1.262 ** 198.3898 105.7806 15.5465 92.6091 50.376 1.838 *** 106.9202 97.5120 23.3197 -45.0315 47.283 0.199 * 99.4759 97.5120 23.3197 19640 47.283 <t< td=""></t<></td> | Dependent Predicted Std Error Residual Std Error Student Residual Residual Residual Std Error Student Residual Residual Std Error Student Std Error Stdent Std Error Student Std Error Stdent Std Error Student Std Error Stdent Std Error Std Std Error Stdent Std Erro | Variable Value Mean Predict Residual Residual 158.4964 122.3180 19.0405 36.1785 49.162 0.736 * 119.5232 122.3180 19.0405 -2.7948 49.162 -0.0568 198.4892 122.3180 19.0405 76.1712 49.162 1.549 *** 98.3567 114.0493 13.4636 -15.6926 50.973 -0.308 *** 88.3234 122.3180 19.0405 -33.9945 49.162 -0.691 * ** 122.2845 122.3180 19.0405 -0.0334 49.162 -0.457 ** 60.2688 122.3180 19.0405 -22.4611 49.162 -0.457 ** 60.2688 122.3180 19.0405 -62.0491 49.162 -1.262 ** 198.3898 105.7806 15.5465 92.6091 50.376 1.838 *** 106.9202 97.5120 23.3197 -45.0315 47.283 0.199 * 99.4759 97.5120 23.3197 19640 47.283 <t< td=""></t<> |

Sum of Residuals Sum of Squared Residuals 38913 Predicted Residual SS (PRESS) 48950

## ----- SUMMARY REPORT -----

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=Cmax

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source Model 1 8057.83696 8057.83696 0.45 0.5149
Error 14 252708 18051
Corrected Total 15 260766

> Root MSE 134.35239 R-Square 0.0309 Dependent Mean 303.87500 Adj R-Sq -0.0383 Coeff Var 44.21305

#### Parameter Estimates

Variable DF Parameter Standard t Value Pr > |t| 95% Confidence Limits
Intercept 1 186.89130 178.28262 1.05 0.3123 -195.48688 569.26948 indiv 1 18.71739 28.01441 0.67 0.5149 -41.36754 78.80233

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=Cmax

#### Output Statistics

| | | | Outp | out Statis | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted Value | Error<br>Predict | Residual | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 159.0000 | 280.4783 | 48.5224 | -121.4783 | 125.3 | -0.970 | * | | 0.071 |
| 2 | 350.0000 | 280.4783 | 48.5224 | 69.5217 | 125.3 | 0.555 | | * | 0.023 |
| 3 | 125.0000 | 280.4783 | 48.5224 | -155.4783 | 125.3 | -1.241 | ** | | 0.116 |
| 4 | 518.0000 | 299.1957 | 34.3105 | 218.8043 | 129.9 | 1.684 | | *** | 0.099 |
| 5 | 255.0000 | 280.4783 | 48.5224 | -25.4783 | 125.3 | -0.203 | | | 0.003 |
| 6 | 258.0000 | 280.4783 | 48.5224 | -22.4783 | 125.3 | -0.179 | | | 0.002 |
| 7 | 220.0000 | 280.4783 | 48.5224 | -60.4783 | 125.3 | -0.483 | | | 0.017 |
| 8 | 416.0000 | 280.4783 | 48.5224 | 135.5217 | 125.3 | 1.082 | | * * | 0.088 |
| 9 | 207.0000 | 317.9130 | 39.6184 | -110.9130 | 128.4 | -0.864 | * | | 0.036 |
| 10 | 259.0000 | 336.6304 | 59.4275 | -77.6304 | 120.5 | -0.644 | * | | 0.050 |
| 11 | 388.0000 | 336.6304 | 59.4275 | 51.3696 | 120.5 | 0.426 | | | 0.022 |
| 12 | 221.0000 | 336.6304 | 59.4275 | -115.6304 | 120.5 | -0.960 | * | | 0.112 |
| 13 | 359.0000 | 317.9130 | 39.6184 | 41.0870 | 128.4 | 0.320 | | | 0.005 |
| 14 | 419.0000 | 317.9130 | 39.6184 | 101.0870 | 128.4 | 0.787 | | * | 0.030 |
| 15 | 143.0000 | 317.9130 | 39.6184 | -174.9130 | 128.4 | -1.362 | ** | | 0.088 |
| 16 | 565.0000 | 317.9130 | 39.6184 | 247.0870 | 128.4 | 1.925 | | *** | 0.176 |
| 17 | 199.0000 | | | | | | | | |
| 18 | 307.0000 | | | | | | | | |
| 19 | 216.0000 | | | | | | | | |
| 20 | 270.0000 | | | | | | | | |
| 21 | 189.0000 | | | | | | | | |
| 22 | 288.0000 | | | | | | | | |
| 23 | 149.0000 | | | | | | | | |
| 24 | 192.0000 | | | | | | | | |

Sum of Residuals 0 Sum of Squared Residuals 252708 Predicted Residual SS (PRESS) 316352 Algorithme Pharma

#### CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=LambdaZ

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

Analysis of Variance

DF Sum of Mean F Value Pr > F Source

Squares Square

Model

Error 14 0.01398 0.00099868 Corrected Total 15 0.01748

Root MSE 0.03160 R-Square 0.2000 Dependent Mean 0.10757 Adj R-Sq 0.1428

Coeff Var 29.37706

#### Parameter Estimates

Variable DF Parameter Standard t Value Pr > |t| 95% Estimate Error Confidence Limits

Intercept 1 0.18461 0.04194 4.40 0.0006 0.09467 0.27456 indiv 1 -0.01233 0.00659 -1.87 0.0824 -0.02646 0.00181

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

### NAME OF FORMER VARIABLE=LambdaZ

#### Output Statistics

| 01 | | D 1' ' 1 | - | out Statis | | G. 1 . | | 0.1.0 | a 1. |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2 | 0 1 2 | Cook's<br>D |
| 1 | 0.0999 | 0.1230 | 0.0114 | -0.0231 | | | * | 1 1 | 0.046 |
| | | | | | | | ** | !!! | |
| 2 | 0.0872 | 0.1230 | 0.0114 | -0.0358 | | | . ** | !!! | 0.110 |
| 3 | 0.1578 | 0.1230 | 0.0114 | 0.0348 | 0.0295 | | | ** | 0.105 |
| 4 | 0.1939 | 0.1107 | 0.008070 | 0.0832 | 0.0306 | 2.724 | | **** | 0.259 |
| 5 | 0.1032 | 0.1230 | 0.0114 | -0.0197 | 0.0295 | -0.670 | * | | 0.034 |
| 6 | 0.1643 | 0.1230 | 0.0114 | 0.0413 | 0.0295 | 1.401 | | ** | 0.147 |
| 7 | 0.0981 | 0.1230 | 0.0114 | -0.0249 | 0.0295 | -0.844 | * | | 0.053 |
| 8 | 0.1020 | 0.1230 | 0.0114 | -0.0210 | 0.0295 | -0.713 | * | | 0.038 |
| 9 | 0.1045 | 0.0983 | 0.009319 | 0.006156 | 0.0302 | 0.204 | | | 0.002 |
| 10 | 0.0943 | 0.0860 | 0.0140 | 0.008283 | 0.0283 | 0.292 | | | 0.010 |
| 11 | 0.0777 | 0.0860 | 0.0140 | -0.008316 | 0.0283 | -0.293 | | | 0.010 |
| 12 | 0.0727 | 0.0860 | 0.0140 | -0.0133 | 0.0283 | -0.470 | | | 0.027 |
| 13 | 0.0892 | 0.0983 | 0.009319 | -0.009175 | 0.0302 | -0.304 | | | 0.004 |
| 14 | 0.0799 | 0.0983 | 0.009319 | -0.0184 | 0.0302 | -0.609 | * | | 0.018 |
| 15 | 0.1053 | 0.0983 | 0.009319 | 0.006991 | 0.0302 | 0.232 | | | 0.003 |
| 16 | 0.0912 | 0.0983 | 0.009319 | -0.007169 | 0.0302 | -0.237 | İ | | 0.003 |
| 17 | 0.1274 | | | | | | | | |
| 18 | 0.1519 | | | | | | | | |
| 19 | 0.1231 | | | | | | | | |
| 20 | 0.1469 | | | | | | | | |
| 21 | 0.1513 | | | | | | | | |
| 22 | 0.1428 | | | | | | | | |
| 23 | 0.1299 | | | | | | | | |
| 24 | 0.1211 | | | | | | | | |

Sum of Residuals 0 Sum of Squared Residuals 0.01398 Predicted Residual SS (PRESS) 0.01726 Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=RkTmax

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

Analysis of Variance

DF Sum of Mean F Value Pr > F Source

Squares Square

1 152.63315 152.63315 4.91 0.0437 Model

Error 14 434.80435 31.05745

Corrected Total 15 587.43750

Root MSE 5.57292 R-Square 0.2598 Dependent Mean 9.68750 Adj R-Sq 0.2070

Coeff Var 57.52693

#### Parameter Estimates

Variable DF Parameter Standard t Value Pr > |t| 95% Estimate Error Confidence Limits

Intercept 1 25.78804 7.39514 3.49 0.0036 9.92704 41.64905 indiv 1 -2.57609 1.16203 -2.22 0.0437 -5.06840 -0.08377

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

# Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

### NAME OF FORMER VARIABLE=RkTmax

#### Output Statistics

| | | | - | ul Statis | | a | | | ~ 1. |
|---|---|---|---|---|---|---|---|---|---|
| Obs | _ | Predicted | Std Error<br>Mean Predict | | Std Error | | -2-1 | 0 1 2 | Cook's |
| | Variable | | | | Residual | | | | D |
| 1 | 14.0000 | 12.9076 | 2.0127 | 1.0924 | 5.197 | 0.210 | | | 0.003 |
| 2 | 2.0000 | 12.9076 | 2.0127 | -10.9076 | 5.197 | -2.099 | **** | | 0.330 |
| 3 | 14.0000 | 12.9076 | 2.0127 | 1.0924 | 5.197 | 0.210 | | | 0.003 |
| 4 | 2.0000 | 10.3315 | 1.4232 | -8.3315 | 5.388 | -1.546 | *** | | 0.083 |
| 5 | 18.0000 | 12.9076 | 2.0127 | 5.0924 | 5.197 | 0.980 | | * | 0.072 |
| 6 | 18.0000 | 12.9076 | 2.0127 | 5.0924 | 5.197 | 0.980 | | * | 0.072 |
| 7 | 21.5000 | 12.9076 | 2.0127 | 8.5924 | 5.197 | 1.653 | | *** | 0.205 |
| 8 | 8.0000 | 12.9076 | 2.0127 | -4.9076 | 5.197 | -0.944 | * | | 0.067 |
| 9 | 5.5000 | 7.7554 | 1.6434 | -2.2554 | 5.325 | -0.424 | | | 0.009 |
| 10 | 5.5000 | 5.1793 | 2.4650 | 0.3207 | 4.998 | 0.0642 | | | 0.001 |
| 11 | 8.0000 | 5.1793 | 2.4650 | 2.8207 | 4.998 | 0.564 | | * | 0.039 |
| 12 | 4.0000 | 5.1793 | 2.4650 | -1.1793 | 4.998 | -0.236 | | | 0.007 |
| 13 | 14.0000 | 7.7554 | 1.6434 | 6.2446 | 5.325 | 1.173 | | ** | 0.065 |
| 14 | 2.0000 | 7.7554 | 1.6434 | -5.7554 | 5.325 | -1.081 | ** | | 0.056 |
| 15 | 10.5000 | 7.7554 | 1.6434 | 2.7446 | 5.325 | 0.515 | | * | 0.013 |
| 16 | 8.0000 | 7.7554 | 1.6434 | 0.2446 | 5.325 | 0.0459 | | | 0.000 |
| 17 | 23.5000 | | | | | | | | |
| 18 | 10.5000 | | | | | | | | |
| 19 | 14.0000 | | | | | | | | |
| 20 | 14.0000 | | | | | | | | |
| 21 | 18.0000 | | | | | | | | |
| 22 | 20.0000 | | | | | | | | |
| 23 | 21.5000 | | | | | | | | |
| 24 | 23.5000 | | | | | | | | |

Sum of Residuals 0 Sum of Squared Residuals 434.80435 Predicted Residual SS (PRESS) 554.34864 Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=Vz F

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

1 17826 17826 0.08 0.7823 Model

14 3145409 224672 Error

Corrected Total 15 3163235

Root MSE 473.99586 R-Square 0.0056 Dependent Mean 1067.91793 Adj R-Sq -0.0654

Coeff Var 44.38505

Variable DF Parameter Standard t Value Pr > |t| 95%
Confidence Limits Estimate Error Confidence Limits
Intercept 1 893.92274 628.98190 1.42 0.1771 -455.10926 2242.95473

indiv 1 27.83923 98.83497 0.28 0.7823 -184.14070 239.81916
## Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=Vz F

## Output Statistics

| Obs | Dependent | Predicted | Std Error | | Std Error | Student | -2-1 | 0 1 2 | Cook's |
|---|---|---|---|---|---|---|---|---|---|
| | Variable | Value | Mean Predict | | Residual | Residual | | | D |
| 1 | 1586 | 1033 | 171.1872 | 553.1365 | 442.0 | 1.251 | | ** | 0.117 |
| 2 | 1370 | 1033 | 171.1872 | 337.0904 | 442.0 | 0.763 | | * | 0.044 |
| 3 | 1258 | 1033 | 171.1872 | 224.5945 | 442.0 | 0.508 | | * | 0.019 |
| 4 | 507.2843 | 1061 | 121.0476 | -553.6738 | 458.3 | -1.208 | ** | | 0.051 |
| 5 | 855.4525 | 1033 | 171.1872 | -177.6664 | 442.0 | -0.402 | | | 0.012 |
| 6 | 744.3830 | 1033 | 171.1872 | -288.7359 | 442.0 | -0.653 | * | | 0.032 |
| 7 | 1018 | 1033 | 171.1872 | -15.2366 | 442.0 | -0.0345 | | | 0.000 |
| 8 | 590.9625 | 1033 | 171.1872 | -442.1564 | 442.0 | -1.000 | ** | | 0.075 |
| 9 | 1899 | 1089 | 139.7738 | 809.9520 | 452.9 | 1.788 | | *** | 0.152 |
| 10 | 1134 | 1117 | 209.6606 | 17.3665 | 425.1 | 0.0409 | | | 0.000 |
| 11 | 675.5488 | 1117 | 209.6606 | -441.0878 | 425.1 | -1.038 | ** | | 0.131 |
| 12 | 1369 | 1117 | 209.6606 | 252.0998 | 425.1 | 0.593 | | * | 0.043 |
| 13 | 806.7430 | 1089 | 139.7738 | -282.0544 | 452.9 | -0.623 | * | | 0.018 |
| 14 | 774.0737 | 1089 | 139.7738 | -314.7236 | 452.9 | -0.695 | * | | 0.023 |
| 15 | 1925 | 1089 | 139.7738 | 836.4027 | 452.9 | 1.847 | | *** | 0.162 |
| 16 | 573.4898 | 1089 | 139.7738 | -515.3075 | 452.9 | -1.138 | ** | | 0.062 |
| 17 | 816.6712 | | | | | | | | |
| 18 | 703.8423 | | | | | | | | |
| 19 | 887.4080 | | | | | | | | |
| 20 | 770.4741 | | | | | | | | |
| 21 | 1168 | | | | | | | | |
| 22 | 652.5078 | | | | | | | | |
| 23 | 1680 | | | | | | | | |
| 24 | 957.1601 | | | | | | | | |

Sum of Residuals Sum of Squared Residuals 3145409 Predicted Residual SS (PRESS) 3941589

## Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1AUCT

Number of Observations Read Number of Observations Used 16
Number of Observations with Missing Values 8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F Squares Square

1 0.17827 0.17827 0.85 0.3725 Model

Error 14 2.94011 0.21001 Corrected Total 15 3.11839

Root MSE 0.45827 R-Square 0.0572 Dependent Mean 7.55526 Adj R-Sq -0.0102 Coeff Var 6.06552

| Variable | DF : | Parameter | Standard t | Value | Pr > | t | 95% |
|---|---|---|---|---|---|---|---|
| | | Estimate | Error | | | | Confidence |
| | | | | | | | Limits |
| Intercept | 1 | 7.00502 | 0.60811 | 11.52 | < .00 | 001 | 5.70075 8.30928 |
| indiv | 1 | 0.08804 | 0.09556 | 0.92 | 0.37 | 725 | -0.11691 0.29299 |

## 

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

## NAME OF FORMER VARIABLE=1AUCT

#### Output Statistics

| | | | - | ut Statis | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| | | | | | | | 1 | | |
| 1 | 7.1142 | 7.4452 | 0.1655 | -0.3310 | 0.427 | -0.775 | * | | 0.045 |
| 2 | 7.3961 | 7.4452 | 0.1655 | -0.0491 | 0.427 | -0.115 | | | 0.001 |
| 3 | 6.8861 | 7.4452 | 0.1655 | -0.5591 | 0.427 | -1.308 | ** | | 0.128 |
| 4 | 7.6107 | 7.5333 | 0.1170 | 0.0775 | 0.443 | 0.175 | | | 0.001 |
| 5 | 7.7018 | 7.4452 | 0.1655 | 0.2566 | 0.427 | 0.600 | | * | 0.027 |
| 6 | 7.3802 | 7.4452 | 0.1655 | -0.0650 | 0.427 | -0.152 | | | 0.002 |
| 7 | 7.5766 | 7.4452 | 0.1655 | 0.1314 | 0.427 | 0.307 | | | 0.007 |
| 8 | 8.0799 | 7.4452 | 0.1655 | 0.6347 | 0.427 | 1.485 | | ** | 0.165 |
| 9 | 6.8675 | 7.6213 | 0.1351 | -0.7538 | 0.438 | -1.722 | *** | | 0.141 |
| 10 | 7.5126 | 7.7093 | 0.2027 | -0.1967 | 0.411 | -0.479 | | | 0.028 |
| 11 | 8.1887 | 7.7093 | 0.2027 | 0.4794 | 0.411 | 1.166 | | ** | 0.165 |
| 12 | 7.5410 | 7.7093 | 0.2027 | -0.1683 | 0.411 | -0.409 | | | 0.020 |
| 13 | 7.8972 | 7.6213 | 0.1351 | 0.2759 | 0.438 | 0.630 | | * | 0.019 |
| 14 | 8.0381 | 7.6213 | 0.1351 | 0.4168 | 0.438 | 0.952 | | * | 0.043 |
| 15 | 6.8784 | 7.6213 | 0.1351 | -0.7429 | 0.438 | -1.696 | *** | | 0.137 |
| 16 | 8.2150 | 7.6213 | 0.1351 | 0.5937 | 0.438 | 1.356 | | ** | 0.088 |
| 17 | 7.5507 | | | | | | | | |
| 18 | 7.5300 | | | | | | | | |
| 19 | 7.5023 | | | | | | | | |
| 20 | 7.4556 | | | | | | | | |
| 21 | 7.0143 | | | | | | | | |
| 22 | 7.6667 | | | | | | | | |
| 23 | 6.7872 | | | | | | | | |
| 24 | 7.4421 | | | | | | | | |

Sum of Residuals Sum of Squared Residuals 2.94011 Predicted Residual SS (PRESS) 3.74168

## Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1AUCinf

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

1 0.20718 0.20718 0.98 0.3394 Model

Error 14 2.96475 0.21177

Corrected Total 15 3.17193

Root MSE 0.46018 R-Square 0.0653 Dependent Mean 7.58666 Adj R-Sq -0.0014

Coeff Var 6.06568

| Variable | DF I | Parameter | Standard t | Value : | Pr > t | 95% |
|---|---|---|---|---|---|---|
| | | Estimate | Error | | | Confidence |
| | | | | | | Limits |
| Intercept | 1 | 6.99347 | 0.61065 | 11.45 | <.0001 | 5.68375 8.30319 |
| indiv | 1 | 0.09491 | 0.09595 | 0.99 | 0.3394 | -0.11089 0.30071 |

## Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

## NAME OF FORMER VARIABLE=1AUCinf

#### Output Statistics

| Obs | Donondont | Drodiatod | - | ut Statis | Std Error | Ctudont | 2 1 | 0 1 2 | Cook's |
|---|---|---|---|---|---|---|---|---|---|
| ODS | Variable | | Mean Predict | | Residual | | -2-1 | 0 1 2 | D D |
| 1 | 7.1403 | 7.4680 | 0.1662 | -0.3277 | 0.429 | -0.764 | * | | 0.044 |
| 2 | 7.4226 | 7.4680 | 0.1662 | -0.0455 | 0.429 | -0.106 | i | | 0.001 |
| 3 | 6.9153 | 7.4680 | 0.1662 | | 0.429 | -1.288 | ** | ' ' | 0.124 |
| 4 | 7.6175 | 7.5629 | 0.1175 | | 0.445 | 0.123 | i | ' '<br> | 0.001 |
| 5 | 7.7251 | | 0.1662 | | 0.429 | 0.599 | i | * | 0.027 |
| 6 | 7.3997 | 7.4680 | 0.1662 | | 0.429 | -0.159 | i | ' '<br> | 0.002 |
| 7 | 7.6023 | 7.4680 | 0.1662 | | 0.429 | 0.313 | i | | 0.007 |
| 8 | 8.1073 | 7.4680 | 0.1662 | | 0.429 | 1.490 | i | ** | 0.166 |
| 9 | 6.9158 | 7.6578 | 0.1357 | -0.7420 | 0.440 | -1.687 | *** | | 0.136 |
| 10 | 7.5340 | 7.7527 | 0.2036 | -0.2188 | 0.413 | -0.530 | * | | 0.034 |
| 11 | 8.2456 | 7.7527 | 0.2036 | 0.4929 | 0.413 | 1.194 | i | ** | 0.173 |
| 12 | 7.6062 | 7.7527 | 0.2036 | -0.1466 | 0.413 | -0.355 | i | | 0.015 |
| 13 | 7.9305 | 7.6578 | 0.1357 | 0.2726 | 0.440 | 0.620 | i | * | 0.018 |
| 14 | 8.0808 | 7.6578 | 0.1357 | 0.4230 | 0.440 | 0.962 | İ | * | 0.044 |
| 15 | 6.8940 | 7.6578 | 0.1357 | -0.7638 | 0.440 | -1.737 | *** | İ | 0.144 |
| 16 | 8.2495 | 7.6578 | 0.1357 | 0.5916 | 0.440 | 1.345 | İ | ** | 0.086 |
| 17 | 7.5616 | | | | | | | | |
| 18 | 7.5339 | | | | | | | | |
| 19 | 7.5129 | | | | | | | | |
| 20 | 7.4773 | | | | | | | | |
| 21 | 7.0311 | | | | | | | | |
| 22 | 7.6717 | | | | | | | | |
| 23 | 6.8206 | | | | | | | | |
| 24 | 7.4529 | | | | | | | | |

Sum of Residuals Sum of Squared Residuals 2.96475 Predicted Residual SS (PRESS) 3.77644

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1CLF

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F Squares Square

1 0.20718 0.20718 0.98 0.3394 Model

Error 14 2.96475 0.21177 Corrected Total 15 3.17193

Root MSE 0.46018 R-Square 0.0653 Dependent Mean 4.61942 Adj R-Sq -0.0014 Coeff Var 9.96191

| Variable | DF | Parameter | Standard t | Value F | r > t | 95% |
|---|---|---|---|---|---|---|
| | | Estimate | Error | | | Confidence |
| | | | | | | Limits |
| Intercept | 1 | 5.21260 | 0.61065 | 8.54 | <.0001 | 3.90289 6.52232 |
| indiv | 1 | -0.09491 | 0.09595 | -0.99 | 0.3394 | -0.30071 0.11089 |

# Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1CLF

#### Output Statistics

| | | | - | ul Statis | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | | | | | Std Error | | -2-1 | 0 1 2 | Cook's |
| | Variable | Value | Mean Predict | | Residual | Residual | | | D |
| 1 | 5.0657 | 4.7381 | 0.1662 | 0.3277 | 0.429 | 0.764 | | * | 0.044 |
| 2 | 4.7835 | 4.7381 | 0.1662 | 0.0455 | 0.429 | 0.106 | | | 0.001 |
| 3 | 5.2907 | 4.7381 | 0.1662 | 0.5527 | 0.429 | 1.288 | | ** | 0.124 |
| 4 | 4.5886 | 4.6431 | 0.1175 | -0.0545 | 0.445 | -0.123 | | | 0.001 |
| 5 | 4.4810 | 4.7381 | 0.1662 | -0.2570 | 0.429 | -0.599 | * | | 0.027 |
| 6 | 4.8064 | 4.7381 | 0.1662 | 0.0683 | 0.429 | 0.159 | | | 0.002 |
| 7 | 4.6037 | 4.7381 | 0.1662 | -0.1343 | 0.429 | -0.313 | | | 0.007 |
| 8 | 4.0988 | 4.7381 | 0.1662 | -0.6392 | 0.429 | -1.490 | ** | | 0.166 |
| 9 | 5.2902 | 4.5482 | 0.1357 | 0.7420 | 0.440 | 1.687 | 1 | *** | 0.136 |
| 10 | 4.6721 | 4.4533 | 0.2036 | 0.2188 | 0.413 | 0.530 | | * | 0.034 |
| 11 | 3.9604 | 4.4533 | 0.2036 | -0.4929 | 0.413 | -1.194 | ** | | 0.173 |
| 12 | 4.5999 | 4.4533 | 0.2036 | 0.1466 | 0.413 | 0.355 | | | 0.015 |
| 13 | 4.2756 | 4.5482 | 0.1357 | -0.2726 | 0.440 | -0.620 | * | | 0.018 |
| 14 | 4.1253 | 4.5482 | 0.1357 | -0.4230 | 0.440 | -0.962 | * | | 0.044 |
| 15 | 5.3120 | 4.5482 | 0.1357 | 0.7638 | 0.440 | 1.737 | | *** | 0.144 |
| 16 | 3.9566 | 4.5482 | 0.1357 | -0.5916 | 0.440 | -1.345 | ** | | 0.086 |
| 17 | 4.6445 | | | | | | | | |
| 18 | 4.6722 | | | | | | | | |
| 19 | 4.6932 | | | | | | | | |
| 20 | 4.7288 | | | | | | | | |
| 21 | 5.1750 | | | | | | | | |
| 22 | 4.5344 | | | | | | | | |
| 23 | 5.3855 | | | | | | | | |
| 24 | 4.7532 | | | | | | | | |

Sum of Residuals 0 Sum of Squared Residuals 2.96475 Predicted Residual SS (PRESS) 3.77644 Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1Cmax

Number of Observations Read Number of Observations Used Number of Observations with Missing Values 8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

1 0.11320 0.11320 0.54 0.4751 Model

Error 14 2.94268 0.21019 Corrected Total 15 3.05588

Root MSE 0.45847 R-Square 0.0370 Dependent Mean 5.62458 Adj R-Sq -0.0317

Coeff Var 8.15113

| Variable | DF 1 | Parameter | Standard t | Value F | r > t | 95% |
|---|---|---|---|---|---|---|
| | | Estimate | Error | | | Confidence |
| | | | | | | Limits |
| Intercept | 1 | 5.18611 | 0.60837 | 8.52 | <.0001 | 3.88127 6.49094 |
| indiv | 1 | 0.07016 | 0.09560 | 0.73 | 0.4751 | -0.13488 0.27519 |

## Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

## NAME OF FORMER VARIABLE=1Cmax

#### Output Statistics

| | | | Outp | ut Statis | SCICS | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Error<br>Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 5.0689 | 5.5369 | 0.1656 | -0.4680 | 0.428 | -1.095 | ** | | 0.090 |
| 2 | 5.8579 | 5.5369 | 0.1656 | 0.3211 | 0.428 | 0.751 | | * | 0.042 |
| 3 | 4.8283 | 5.5369 | 0.1656 | -0.7086 | 0.428 | -1.657 | *** | | 0.206 |
| 4 | 6.2500 | 5.6070 | 0.1171 | 0.6429 | 0.443 | 1.450 | | ** | 0.073 |
| 5 | 5.5413 | 5.5369 | 0.1656 | 0.004380 | 0.428 | 0.0102 | | | 0.000 |
| 6 | 5.5530 | 5.5369 | 0.1656 | 0.0161 | 0.428 | 0.0376 | | | 0.000 |
| 7 | 5.3936 | 5.5369 | 0.1656 | -0.1433 | 0.428 | -0.335 | | | 0.008 |
| 8 | 6.0307 | 5.5369 | 0.1656 | 0.4938 | 0.428 | 1.155 | | ** | 0.100 |
| 9 | 5.3327 | 5.6772 | 0.1352 | -0.3445 | 0.438 | -0.786 | * | | 0.029 |
| 10 | 5.5568 | 5.7473 | 0.2028 | -0.1905 | 0.411 | -0.463 | | | 0.026 |
| 11 | 5.9610 | 5.7473 | 0.2028 | 0.2137 | 0.411 | 0.520 | | * | 0.033 |
| 12 | 5.3982 | 5.7473 | 0.2028 | -0.3492 | 0.411 | -0.849 | * | | 0.088 |
| 13 | 5.8833 | 5.6772 | 0.1352 | 0.2061 | 0.438 | 0.471 | | | 0.011 |
| 14 | 6.0379 | 5.6772 | 0.1352 | 0.3607 | 0.438 | 0.823 | | * | 0.032 |
| 15 | 4.9628 | 5.6772 | 0.1352 | -0.7143 | 0.438 | -1.631 | *** | | 0.127 |
| 16 | 6.3368 | 5.6772 | 0.1352 | 0.6596 | 0.438 | 1.506 | | *** | 0.108 |
| 17 | 5.2933 | | | | | | | | |
| 18 | 5.7268 | | | | | | | | |
| 19 | 5.3753 | | | | | | | | |
| 20 | 5.5984 | | | | | | | | |
| 21 | 5.2417 | | | | | | | | |
| 22 | 5.6630 | | | | | | | | |
| 23 | 5.0039 | | | | | | | | |
| 24 | 5.2575 | | | | | | | | |

Sum of Residuals 0
Sum of Squared Residuals 2.94268
Predicted Residual SS (PRESS) 3.71153

## Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure
Model: MODEL1
Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1LambdaZ

Number of Observations Read 24
Number of Observations Used 16
Number of Observations with Missing Values 8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

Model 1 0.28942 0.28942 4.76 0.0466

Error 14 0.85103 0.06079

Corrected Total 15 1.14045

Root MSE 0.24655 R-Square 0.2538 Dependent Mean -2.26860 Adj R-Sq 0.2005

Coeff Var -10.86800

#### Parameter Estimates

Variable DF Parameter Standard t Value Pr > |t| 95%
Estimate Error Confidence
Limits

Intercept 1 -1.56749 0.32717 -4.79 0.0003 -2.26920 -0.86579 indiv 1 -0.11218 0.05141 -2.18 0.0466 -0.22244 -0.00191

## Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=lLambdaZ

#### Output Statistics

| | | | _ | ut btatis | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | -2.3034 | | 0.0890 | | | | * | | 0.043 |
| 2 | -2.4392 | -2.1284 | 0.0890 | | 0.230 | | ** | | 0.137 |
| | | | | | | | "" | <br> ** | |
| 3 | -1.8463 | -2.1284 | 0.0890 | | 0.230 | | 1 | | 0.113 |
| 4 | -1.6405 | -2.2406 | 0.0630 | | 0.238 | | ! | **** | 0.221 |
| 5 | -2.2706 | -2.1284 | 0.0890 | -0.1422 | 0.230 | -0.619 | * | | 0.029 |
| 6 | -1.8062 | -2.1284 | 0.0890 | 0.3222 | 0.230 | 1.401 | | ** | 0.147 |
| 7 | -2.3217 | -2.1284 | 0.0890 | -0.1934 | 0.230 | -0.841 | * | | 0.053 |
| 8 | -2.2829 | -2.1284 | 0.0890 | -0.1546 | 0.230 | -0.672 | * | | 0.034 |
| 9 | -2.2587 | -2.3527 | 0.0727 | 0.0940 | 0.236 | 0.399 | | | 0.008 |
| 10 | -2.3614 | -2.4649 | 0.1091 | 0.1035 | 0.221 | 0.468 | | | 0.027 |
| 11 | -2.5551 | -2.4649 | 0.1091 | -0.0902 | 0.221 | -0.408 | | | 0.020 |
| 12 | -2.6217 | -2.4649 | 0.1091 | -0.1568 | 0.221 | -0.709 | * | | 0.061 |
| 13 | -2.4174 | -2.3527 | 0.0727 | -0.0647 | 0.236 | -0.274 | | | 0.004 |
| 14 | -2.5264 | -2.3527 | 0.0727 | -0.1737 | 0.236 | -0.737 | * | | 0.026 |
| 15 | -2.2508 | -2.3527 | 0.0727 | 0.1020 | 0.236 | 0.433 | | | 0.009 |
| 16 | -2.3951 | -2.3527 | 0.0727 | -0.0424 | 0.236 | -0.180 | | | 0.002 |
| 17 | -2.0608 | | | | | | | | |
| 18 | -1.8844 | | | | | | | | |
| 19 | -2.0951 | | | | | | | | |
| 20 | -1.9182 | | | | | | | | |
| 21 | -1.8884 | | | | | | | | |
| 22 | -1.9465 | | | | | | | | |
| 23 | -2.0413 | | | | | | | | |
| 24 | -2.1108 | | | | | | | | |

Sum of Residuals Sum of Squared Residuals 0.85103 Predicted Residual SS (PRESS) 1.06423

## Regression Analysis of Individual Child-Pugh Scores at Baseline

----- SUMMARY REPORT -----

The REG Procedure
Model: MODEL1
Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1Vz F

Number of Observations Read 24
Number of Observations Used 16
Number of Observations with Missing Values 8

#### Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

Model 1 0.00686 0.00686 0.04 0.8539

Error 14 2.72991 0.19499

Corrected Total 15 2.73676

Root MSE 0.44158 R-Square 0.0025 Dependent Mean 6.88801 Adj R-Sq -0.0687 Coeff Var 6.41085

#### Parameter Estimates

Variable DF Parameter Standard t Value Pr > |t| 95%
Estimate Error Confidence
Limits

Intercept 1 6.78010 0.58597 11.57 <.0001 5.52332 8.03687
indiv 1 0.01727 0.09208 0.19 0.8539 -0.18022 0.21475</pre>

# Regression Analysis of Individual Child-Pugh Scores at Baseline ----- SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1Vz F

## Output Statistics

| Obs | Dependent | Predicted | _ | Residual | Std Error | Student | -2-1 | 0 1 2 | Cook's |
|---|---|---|---|---|---|---|---|---|---|
| | Variable | Value | Mean Predict | | Residual | Residual | | | D |
| 1 | 7.3691 | 6.8664 | 0.1595 | 0.5027 | 0.412 | 1.221 | | ** | 0.112 |
| 2 | 7.2227 | 6.8664 | 0.1595 | 0.3563 | 0.412 | 0.865 | | * | 0.056 |
| 3 | 7.1371 | 6.8664 | 0.1595 | 0.2706 | 0.412 | 0.657 | | * | 0.032 |
| 4 | 6.2291 | 6.8837 | 0.1128 | -0.6546 | 0.427 | -1.533 | *** | | 0.082 |
| 5 | 6.7516 | 6.8664 | 0.1595 | -0.1148 | 0.412 | -0.279 | | | 0.006 |
| 6 | 6.6126 | 6.8664 | 0.1595 | -0.2539 | 0.412 | -0.617 | * | | 0.029 |
| 7 | 6.9255 | 6.8664 | 0.1595 | 0.0590 | 0.412 | 0.143 | | | 0.002 |
| 8 | 6.3818 | 6.8664 | 0.1595 | -0.4847 | 0.412 | -1.177 | ** | | 0.104 |
| 9 | 7.5490 | 6.9010 | 0.1302 | 0.6480 | 0.422 | 1.536 | | *** | 0.112 |
| 10 | 7.0335 | 6.9182 | 0.1953 | 0.1153 | 0.396 | 0.291 | | | 0.010 |
| 11 | 6.5155 | 6.9182 | 0.1953 | -0.4027 | 0.396 | -1.017 | ** | | 0.126 |
| 12 | 7.2216 | 6.9182 | 0.1953 | 0.3034 | 0.396 | 0.766 | | * | 0.071 |
| 13 | 6.6930 | 6.9010 | 0.1302 | -0.2080 | 0.422 | -0.493 | | | 0.012 |
| 14 | 6.6517 | 6.9010 | 0.1302 | -0.2493 | 0.422 | -0.591 | * | | 0.017 |
| 15 | 7.5628 | 6.9010 | 0.1302 | 0.6618 | 0.422 | 1.569 | | *** | 0.117 |
| 16 | 6.3517 | 6.9010 | 0.1302 | -0.5492 | 0.422 | -1.302 | ** | | 0.081 |
| 17 | 6.7052 | | | | | | | | |
| 18 | 6.5566 | | | | | | | | |
| 19 | 6.7883 | | | | | | | | |
| 20 | 6.6470 | | | | | | | | |
| 21 | 7.0634 | | | | | | | | |
| 22 | 6.4808 | | | | | | | | |
| 23 | 7.4268 | | | | | | | | |
| 24 | 6.8640 | | | | | | | | |

Sum of Residuals 0 Sum of Squared Residuals 2.72991 Predicted Residual SS (PRESS) 3.43815

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=AUCT

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 2 2044534 1022267 1.66 0.2144

21 12944140 616388

Corrected Total 23 14988674

785.10359 R-Square 0.1364 Root MSE Dependent Mean 1947.14710 Adj R-Sq 0.0542

Coeff Var 40.32071

| Variable | DF | Parameter | Standard | t | Value Pr | ^ > | · t | 95% |
|---|---|---|---|---|---|---|---|---|
| | | Estimate | Error | | | | | Confidence Limits |
| Intercept | 1 : | 1643.50654 | 277.57604 | | 5.92 | <. | 0001 | 1066.25558 2220.75751 |
| GrpA | 1 | 213.31383 | 392.55179 | | 0.54 | 0. | 5926 | -603.04231 1029.66998 |
| GrpB | 1 | 697.60783 | 392.55179 | | 1.78 | 0. | 0900 | -118.74831 1513.96398 |

## Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=AUCT

## Output Statistics

| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 1229 | 1857 | 277.5760 | -627.5029 | 734.4 | -0.854 | * | | 0.035 |
| 2 | 1630 | 1857 | 277.5760 | -227.2179 | 734.4 | -0.309 | | | 0.005 |
| 3 | 978.5525 | 1857 | 277.5760 | -878.2679 | 734.4 | -1.196 | ** | | 0.068 |
| 4 | 2020 | 1857 | 277.5760 | 162.9546 | 734.4 | 0.222 | | | 0.002 |
| 5 | 2212 | 1857 | 277.5760 | 355.5051 | 734.4 | 0.484 | | | 0.011 |
| 6 | 1604 | 1857 | 277.5760 | -252.9079 | 734.4 | -0.344 | | | 0.006 |
| 7 | 1952 | 1857 | 277.5760 | 95.1996 | 734.4 | 0.130 | | | 0.001 |
| 8 | 3229 | 1857 | 277.5760 | 1372 | 734.4 | 1.869 | | *** | 0.166 |
| 9 | 960.5133 | 2341 | 277.5760 | -1381 | 734.4 | -1.880 | *** | | 0.168 |
| 10 | 1831 | 2341 | 277.5760 | -510.1144 | 734.4 | -0.695 | * | | 0.023 |
| 11 | 3600 | 2341 | 277.5760 | 1259 | 734.4 | 1.714 | | *** | 0.140 |
| 12 | 1884 | 2341 | 277.5760 | -457.3244 | 734.4 | -0.623 | * | | 0.018 |
| 13 | 2690 | 2341 | 277.5760 | 348.6106 | 734.4 | 0.475 | | | 0.011 |
| 14 | 3097 | 2341 | 277.5760 | 755.5406 | 734.4 | 1.029 | | ** | 0.050 |
| 15 | 971.0900 | 2341 | 277.5760 | -1370 | 734.4 | -1.866 | *** | | 0.166 |
| 16 | 3696 | 2341 | 277.5760 | 1355 | 734.4 | 1.845 | | *** | 0.162 |
| 17 | 1902 | 1644 | 277.5760 | 258.5785 | 734.4 | 0.352 | | | 0.006 |
| 18 | 1863 | 1644 | 277.5760 | 219.5410 | 734.4 | 0.299 | | | 0.004 |
| 19 | 1812 | 1644 | 277.5760 | 168.7110 | 734.4 | 0.230 | | | 0.003 |
| 20 | 1729 | 1644 | 277.5760 | 85.9535 | 734.4 | 0.117 | | | 0.001 |
| 21 | 1112 | 1644 | 277.5760 | -531.0890 | 734.4 | -0.723 | * | | 0.025 |
| 22 | 2136 | 1644 | 277.5760 | 492.5518 | 734.4 | 0.671 | | * | 0.021 |
| 23 | 886.3850 | 1644 | 277.5760 | -757.1215 | 734.4 | -1.031 | ** | | 0.051 |
| 24 | 1706 | 1644 | 277.5760 | 62.8750 | 734.4 | 0.0856 | | | 0.000 |

Sum of Residuals 0 Sum of Squared Residuals 12944140 Predicted Residual SS (PRESS) 16906632 ----- SUMMARY REPORT -----Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=AUCT

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 1022267 1.66 0.2144

Denominator 21 616388

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=AUCinf

Number of Observations Read 24 Number of Observations Used 24

## Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 2 2536727 1268364 1.91 0.1728

21 13940255 663822

Corrected Total 23 16476982

Root MSE 814.75252 R-Square 0.1540 Dependent Mean 2001.41149 Adj R-Sq 0.0734

Coeff Var 40.70890

| Variable | DF | Parameter | Standard | t | Value Pi | r | > | t | 95% |
|---|---|---|---|---|---|---|---|---|---|
| | | Estimate | Error | | | | | | Confidence Limits |
| Intercept | 1 3 | 1663.96617 | 288.05852 | | 5.78 | < | .00 | 01 | 1064.91569 2263.01665 |
| GrpA | 1 | 235.71753 | 407.37626 | | 0.58 | 0 | .56 | 90 | -611.46778 1082.90284 |
| GrpB | 1 | 776.61841 | 407.37626 | | 1.91 | 0 | .07 | 04 | -70.56690 1623.80373 |

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

#### The REG Procedure Model: MODEL1 Dependent Variable: Value

## NAME OF FORMER VARIABLE=AUCinf

#### Output Statistics

| Obs | Dependent | | Std Error | Residual | Std Error | | -2-1 | 0 1 2 | Cook's |
|---|---|---|---|---|---|---|---|---|---|
| | Variable | | Mean Predict | | Residual | | | | D |
| 1 | 1262 | 1900 | 288.0585 | -637.8258 | 762.1 | -0.837 | * | | 0.033 |
| 2 | 1673 | 1900 | 288.0585 | -226.3677 | 762.1 | -0.297 | | | 0.004 |
| 3 | 1008 | 1900 | 288.0585 | -892.0720 | 762.1 | -1.170 | ** | | 0.065 |
| 4 | 2033 | 1900 | 288.0585 | 133.7317 | 762.1 | 0.175 | | | 0.001 |
| 5 | 2264 | 1900 | 288.0585 | 364.7209 | 762.1 | 0.479 | | | 0.011 |
| 6 | 1636 | 1900 | 288.0585 | -264.1537 | 762.1 | -0.347 | | | 0.006 |
| 7 | 2003 | 1900 | 288.0585 | 103.1843 | 762.1 | 0.135 | | | 0.001 |
| 8 | 3318 | 1900 | 288.0585 | 1419 | 762.1 | 1.862 | | *** | 0.165 |
| 9 | 1008 | 2441 | 288.0585 | -1432 | 762.1 | -1.880 | *** | | 0.168 |
| 10 | 1871 | 2441 | 288.0585 | -570.0308 | 762.1 | -0.748 | * | | 0.027 |
| 11 | 3811 | 2441 | 288.0585 | 1370 | 762.1 | 1.798 | | *** | 0.154 |
| 12 | 2011 | 2441 | 288.0585 | -430.0475 | 762.1 | -0.564 | * | | 0.015 |
| 13 | 2781 | 2441 | 288.0585 | 340.1253 | 762.1 | 0.446 | | | 0.009 |
| 14 | 3232 | 2441 | 288.0585 | 791.2447 | 762.1 | 1.038 | | ** | 0.051 |
| 15 | 986.3843 | 2441 | 288.0585 | -1454 | 762.1 | -1.908 | *** | | 0.173 |
| 16 | 3826 | 2441 | 288.0585 | 1385 | 762.1 | 1.817 | | *** | 0.157 |
| 17 | 1923 | 1664 | 288.0585 | 258.9952 | 762.1 | 0.340 | | | 0.005 |
| 18 | 1870 | 1664 | 288.0585 | 206.4075 | 762.1 | 0.271 | | | 0.003 |
| 19 | 1832 | 1664 | 288.0585 | 167.5594 | 762.1 | 0.220 | | | 0.002 |
| 20 | 1767 | 1664 | 288.0585 | 103.4880 | 762.1 | 0.136 | | | 0.001 |
| 21 | 1131 | 1664 | 288.0585 | -532.7030 | 762.1 | -0.699 | * | | 0.023 |
| 22 | 2147 | 1664 | 288.0585 | 482.7817 | 762.1 | 0.633 | | * | 0.019 |
| 23 | 916.5388 | 1664 | 288.0585 | -747.4274 | 762.1 | -0.981 | * | | 0.046 |
| 24 | 1725 | 1664 | 288.0585 | 60.8987 | 762.1 | 0.0799 | | | 0.000 |

Sum of Residuals 0 Sum of Squared Residuals 13940255 Predicted Residual SS (PRESS) 18207680 ----- SUMMARY REPORT -----Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=AUCinf

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 1268364 1.91 0.1728

Denominator 21 663822

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=CL F

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance

DF Sum of Mean Squares Square Mean F Value Pr > F Source

Model 2 2288.42227 1144.21114 0.45 0.6432

Error 21 53315 2538.82052 Corrected Total 23 55604

Root MSE 50.38671 R-Square 0.0412 Dependent Mean 117.88031 Adj R-Sq -0.0502

Coeff Var 42.74396

| Variable | DF Parameter | Standard t | Value Pa | r > t | 9! | 58 |
|---|---|---|---|---|---|---|
| | Estimate | Error | | | Confidence | ce Limits |
| Intercept | 1 129.67669 | 17.81439 | 7.28 | <.0001 | 92.62963 | 166.72375 |
| GrpA | 1 -11.47681 | 25.19335 | -0.46 | 0.6534 | -63.86926 | 40.91564 |
| GrpB | 1 -23.91232 | 25.19335 | -0.95 | 0.3533 | -76.30477 | 28.48013 |

## Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=CL F

## Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 158.4964 | 118.1999 | 17.8144 | 40.2966 | 47.132 | 0.855 | | * | 0.035 |
| 2 | 119.5232 | 118.1999 | 17.8144 | 1.3233 | 47.132 | 0.0281 | | | 0.000 |
| 3 | 198.4892 | 118.1999 | 17.8144 | 80.2893 | 47.132 | 1.703 | | *** | 0.138 |
| 4 | 98.3567 | 118.1999 | 17.8144 | -19.8432 | 47.132 | -0.421 | | | 0.008 |
| 5 | 88.3234 | 118.1999 | 17.8144 | -29.8764 | 47.132 | -0.634 | * | | 0.019 |
| 6 | 122.2845 | 118.1999 | 17.8144 | 4.0846 | 47.132 | 0.0867 | | | 0.000 |
| 7 | 99.8568 | 118.1999 | 17.8144 | -18.3431 | 47.132 | -0.389 | | | 0.007 |
| 8 | 60.2688 | 118.1999 | 17.8144 | -57.9311 | 47.132 | -1.229 | ** | | 0.072 |
| 9 | 198.3898 | 105.7644 | 17.8144 | 92.6254 | 47.132 | 1.965 | | *** | 0.184 |
| 10 | 106.9202 | 105.7644 | 17.8144 | 1.1558 | 47.132 | 0.0245 | | | 0.000 |
| 11 | 52.4805 | 105.7644 | 17.8144 | -53.2839 | 47.132 | -1.131 | ** | | 0.061 |
| 12 | 99.4759 | 105.7644 | 17.8144 | -6.2885 | 47.132 | -0.133 | | | 0.001 |
| 13 | 71.9241 | 105.7644 | 17.8144 | -33.8403 | 47.132 | -0.718 | * | | 0.025 |
| 14 | 61.8845 | 105.7644 | 17.8144 | -43.8799 | 47.132 | -0.931 | * | | 0.041 |
| 15 | 202.7607 | 105.7644 | 17.8144 | 96.9964 | 47.132 | 2.058 | | **** | 0.202 |
| 16 | 52.2793 | 105.7644 | 17.8144 | -53.4850 | 47.132 | -1.135 | ** | | 0.061 |
| 17 | 104.0063 | 129.6767 | 17.8144 | -25.6704 | 47.132 | -0.545 | * | | 0.014 |
| 18 | 106.9305 | 129.6767 | 17.8144 | -22.7462 | 47.132 | -0.483 | | | 0.011 |
| 19 | 109.1986 | 129.6767 | 17.8144 | -20.4781 | 47.132 | -0.434 | | | 0.009 |
| 20 | 113.1571 | 129.6767 | 17.8144 | -16.5196 | 47.132 | -0.350 | | | 0.006 |
| 21 | 176.7935 | 129.6767 | 17.8144 | 47.1168 | 47.132 | 1.000 | | * | 0.048 |
| 22 | 93.1642 | 129.6767 | 17.8144 | -36.5125 | 47.132 | -0.775 | * | | 0.029 |
| 23 | 218.2123 | 129.6767 | 17.8144 | 88.5356 | 47.132 | 1.878 | | *** | 0.168 |
| 24 | 115.9511 | 129.6767 | 17.8144 | -13.7256 | 47.132 | -0.291 | | | 0.004 |

Sum of Residuals 0 Sum of Squared Residuals 53315 Predicted Residual SS (PRESS) 69636 ----- SUMMARY REPORT -----Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=CL\_F

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 1144.21114 0.45 0.6432

Denominator 21 2538.82052

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=Cmax

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance
DF Sum of Mean F Value Pr > F Source

Squares Square

Model 2 36362 18181 1.37 0.2753

21 278164 13246

Corrected Total 23 314526

115.09091 R-Square 0.1156 Root MSE Dependent Mean 278.00000 Adj R-Sq 0.0314

Coeff Var 41.39961

| Variable | DF Parameter Standard t Value Pr > | t 95% |
|-----------|------------------------------------|------------------------|
| | Estimate Error | Confidence Limits |
| Intercept | 1 226.25000 40.69078 5.56 <.00 | 01 141.62889 310.87111 |
| GrpA | 1 61.37500 57.54545 1.07 0.29 | 83 -58.29732 181.04732 |
| GrpB | 1 93.87500 57.54545 1.63 0.11 | 77 -25.79732 213.54732 |

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=Cmax

## Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 159.0000 | 287.6250 | 40.6908 | -128.6250 | 107.7 | -1.195 | ** | | 0.068 |
| 2 | 350.0000 | 287.6250 | 40.6908 | 62.3750 | 107.7 | 0.579 | İ | * | 0.016 |
| 3 | 125.0000 | 287.6250 | 40.6908 | -162.6250 | 107.7 | -1.511 | *** | ĺ | 0.109 |
| 4 | 518.0000 | 287.6250 | 40.6908 | 230.3750 | 107.7 | 2.140 | | **** | 0.218 |
| 5 | 255.0000 | 287.6250 | 40.6908 | -32.6250 | 107.7 | -0.303 | | | 0.004 |
| 6 | 258.0000 | 287.6250 | 40.6908 | -29.6250 | 107.7 | -0.275 | | | 0.004 |
| 7 | 220.0000 | 287.6250 | 40.6908 | -67.6250 | 107.7 | -0.628 | * | | 0.019 |
| 8 | 416.0000 | 287.6250 | 40.6908 | 128.3750 | 107.7 | 1.192 | | ** | 0.068 |
| 9 | 207.0000 | 320.1250 | 40.6908 | -113.1250 | 107.7 | -1.051 | ** | | 0.053 |
| 10 | 259.0000 | 320.1250 | 40.6908 | -61.1250 | 107.7 | -0.568 | * | | 0.015 |
| 11 | 388.0000 | 320.1250 | 40.6908 | 67.8750 | 107.7 | 0.630 | | * | 0.019 |
| 12 | 221.0000 | 320.1250 | 40.6908 | -99.1250 | 107.7 | -0.921 | * | | 0.040 |
| 13 | 359.0000 | 320.1250 | 40.6908 | 38.8750 | 107.7 | 0.361 | | | 0.006 |
| 14 | 419.0000 | 320.1250 | 40.6908 | 98.8750 | 107.7 | 0.918 | | * | 0.040 |
| 15 | 143.0000 | 320.1250 | 40.6908 | -177.1250 | 107.7 | -1.645 | *** | | 0.129 |
| 16 | 565.0000 | 320.1250 | 40.6908 | 244.8750 | 107.7 | 2.275 | | **** | 0.246 |
| 17 | 199.0000 | 226.2500 | 40.6908 | -27.2500 | 107.7 | -0.253 | | | 0.003 |
| 18 | 307.0000 | 226.2500 | 40.6908 | 80.7500 | 107.7 | 0.750 | | * | 0.027 |
| 19 | 216.0000 | 226.2500 | 40.6908 | -10.2500 | 107.7 | -0.0952 | | | 0.000 |
| 20 | 270.0000 | 226.2500 | 40.6908 | 43.7500 | 107.7 | 0.406 | | | 0.008 |
| 21 | 189.0000 | 226.2500 | 40.6908 | -37.2500 | 107.7 | -0.346 | | | 0.006 |
| 22 | 288.0000 | 226.2500 | 40.6908 | 61.7500 | 107.7 | 0.574 | | * | 0.016 |
| 23 | 149.0000 | 226.2500 | 40.6908 | -77.2500 | 107.7 | -0.718 | * | | 0.025 |
| 24 | 192.0000 | 226.2500 | 40.6908 | -34.2500 | 107.7 | -0.318 | | | 0.005 |

Sum of Residuals 0 Sum of Squared Residuals 278164 Predicted Residual SS (PRESS) 363317

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=Cmax

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 18181 1.37 0.2753

Denominator 21 13246

## ----- SUMMARY REPORT -----

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=LambdaZ

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance

DF Sum of Mean F Value Pr > F Source

Squares Square

Model

21 0.01330 0.00063354

Corrected Total 23 0.02318

Root MSE 0.02517 R-Square 0.4259 Dependent Mean 0.11731 Adj R-Sq 0.3713

Coeff Var 21.45595

| Variable | DF: | Parameter: | Standard t | Value P | r > | t | 95 | % |
|---|---|---|---|---|---|---|---|---|
| | Estimate | | Error | | | | Confid | Confidence |
| | | | | | | | Limi | its |
| Intercept | 1 | 0.13679 | 0.00890 | 15.37 | <.00 | 001 | 0.11828 | 0.15529 |
| GrpA | 1 | -0.01098 | 0.01259 | -0.87 | 0.39 | 929 | -0.03715 | 0.01520 |
| GrpB | 1 | -0.04745 | 0.01259 | -3.77 | 0.0 | 011 | -0.07362 | -0.02127 |

## 

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=LambdaZ

## Output Statistics

| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 0.0999 | 0.1258 | 0.008899 | -0.0259 | 0.0235 | -1.100 | ** | | 0.058 |
| 2 | 0.0872 | 0.1258 | 0.008899 | -0.0386 | 0.0235 | -1.639 | *** | | 0.128 |
| 3 | 0.1578 | 0.1258 | 0.008899 | 0.0320 | 0.0235 | 1.360 | | ** | 0.088 |
| 4 | 0.1939 | 0.1258 | 0.008899 | 0.0681 | 0.0235 | 2.892 | | **** | 0.398 |
| 5 | 0.1032 | 0.1258 | 0.008899 | -0.0226 | 0.0235 | -0.958 | * | | 0.044 |
| 6 | 0.1643 | 0.1258 | 0.008899 | 0.0385 | 0.0235 | 1.634 | | *** | 0.127 |
| 7 | 0.0981 | 0.1258 | 0.008899 | -0.0277 | 0.0235 | -1.177 | ** | | 0.066 |
| 8 | 0.1020 | 0.1258 | 0.008899 | -0.0238 | 0.0235 | -1.012 | ** | | 0.049 |
| 9 | 0.1045 | 0.0893 | 0.008899 | 0.0151 | 0.0235 | 0.643 | | * | 0.020 |
| 10 | 0.0943 | 0.0893 | 0.008899 | 0.004947 | 0.0235 | 0.210 | | | 0.002 |
| 11 | 0.0777 | 0.0893 | 0.008899 | -0.0117 | 0.0235 | -0.495 | | | 0.012 |
| 12 | 0.0727 | 0.0893 | 0.008899 | -0.0167 | 0.0235 | -0.708 | * | | 0.024 |
| 13 | 0.0892 | 0.0893 | 0.008899 | -0.000185 | 0.0235 | -0.0079 | | | 0.000 |
| 14 | 0.0799 | 0.0893 | 0.008899 | -0.009393 | 0.0235 | -0.399 | | | 0.008 |
| 15 | 0.1053 | 0.0893 | 0.008899 | 0.0160 | 0.0235 | 0.679 | | * | 0.022 |
| 16 | 0.0912 | 0.0893 | 0.008899 | 0.001821 | 0.0235 | 0.0773 | | | 0.000 |
| 17 | 0.1274 | 0.1368 | 0.008899 | -0.009431 | 0.0235 | -0.401 | | | 0.008 |
| 18 | 0.1519 | 0.1368 | 0.008899 | 0.0151 | 0.0235 | 0.643 | | * | 0.020 |
| 19 | 0.1231 | 0.1368 | 0.008899 | -0.0137 | 0.0235 | -0.583 | * | | 0.016 |
| 20 | 0.1469 | 0.1368 | 0.008899 | 0.0101 | 0.0235 | 0.428 | | | 0.009 |
| 21 | 0.1513 | 0.1368 | 0.008899 | 0.0145 | 0.0235 | 0.617 | | * | 0.018 |
| 22 | 0.1428 | 0.1368 | 0.008899 | 0.005993 | 0.0235 | 0.255 | | | 0.003 |
| 23 | 0.1299 | 0.1368 | 0.008899 | -0.006930 | 0.0235 | -0.294 | | | 0.004 |
| 24 | 0.1211 | 0.1368 | 0.008899 | -0.0156 | 0.0235 | -0.664 | * | | 0.021 |

Sum of Residuals 0 Sum of Squared Residuals 0.01330 Predicted Residual SS (PRESS) 0.01738 CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=LambdaZ

Test test\_FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F

Square

Numerator 2 0.00494 7.79 0.0029

Denominator 21 0.00063354

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=Vz F

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance
DF Sum of Mean F Value Pr > F Source

Squares Square

Model 2 162471 81235 0.44 0.6481

21 3853369 183494

Corrected Total 23 4015840

Root MSE 428.36169 R-Square 0.0405 Dependent Mean 1030.15023 Adj R-Sq -0.0509

Coeff Var 41.58245

| Variable | DF Parameter Standard t | t Value Pr > t | 95% |
|-----------|-------------------------|-----------------|----------------------|
| | Estimate Error | | Confidence Limits |
| Intercept | 1 954.61482 151.44873 | 6.30 <.0001 | 639.65995 1269.56969 |
| GrpA | 1 36.65302 214.18085 | 0.17 0.8658 | -408.76043 482.06648 |
| GrpB | 1 189.95321 214.18085 | 0.89 0.3852 | -255.46025 635.36666 |

# Regression Analysis of Group Child-Pugh Classification at Baseline ------ SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=Vz F

## Output Statistics

| 01 | D | D 22 2 | _ | nuc scacis | | Q+ | 0 1 0 1 | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | kesidual | Std Error<br>Residual | | -2-1 0 1 | l 2 Cook's<br>D |
| 1 | 1586 | 991.2678 | 151.4487 | 594.9876 | 400.7 | 1.485 | ** | 0.105 |
| 2 | 1370 | 991.2678 | 151.4487 | 378.9415 | 400.7 | 0.946 | * | 0.043 |
| 3 | 1258 | 991.2678 | 151.4487 | 266.4455 | 400.7 | 0.665 | * | 0.021 |
| 4 | 507.2843 | 991.2678 | | -483.9835 | 400.7 | | ** | 0.069 |
| 5 | 855.4525 | 991.2678 | | -135.8153 | 400.7 | | i i | 0.005 |
| 6 | 744.3830 | 991.2678 | | -246.8848 | 400.7 | | * | 0.018 |
| 7 | 1018 | 991.2678 | 151.4487 | 26.6144 | 400.7 | | i i | 0.000 |
| 8 | 590.9625 | 991.2678 | | -400.3053 | 400.7 | | * | 0.048 |
| 9 | 1899 | 1145 | 151.4487 | 754.1813 | 400.7 | 1.882 | *** | ! |
| 10 | 1134 | 1145 | 151.4487 | -10.5650 | 400.7 | -0.0264 | i i | 0.000 |
| 11 | 675.5488 | 1145 | | -469.0192 | 400.7 | -1.171 | ** | 0.065 |
| 12 | 1369 | 1145 | 151.4487 | | 400.7 | 0.559 | * | 0.015 |
| 13 | 806.7430 | 1145 | | -337.8251 | 400.7 | | * | 0.013 |
| 14 | 774.0737 | 1145 | | -370.4943 | 400.7 | | * | 0.041 |
| 15 | 1925 | 1145 | 151.4487 | 780.6320 | 400.7 | 1.948 | *** | : |
| 16 | 573.4898 | 1145 | | -571.0782 | 400.7 | -1.425 | ** | 0.097 |
| 17 | 816.6712 | 954.6148 | | -137.9436 | 400.7 | | i i | 0.006 |
| 18 | 703.8423 | 954.6148 | | -250.7725 | 400.7 | | * | 0.019 |
| 19 | 887.4080 | 954.6148 | 151.4487 | | 400.7 | | 1 1 | 0.001 |
| 20 | 770.4741 | 954.6148 | | -184.1407 | 400.7 | -0.460 | i i | 0.010 |
| 21 | 1168 | 954.6148 | 151.4487 | 213.8099 | 400.7 | 0.534 | * | 0.014 |
| 22 | 652.5078 | 954.6148 | | -302.1070 | 400.7 | -0.754 | * | 0.014 |
| 23 | 1680 | 954.6148 | 151.4487 | 725.8154 | 400.7 | 1.811 | *** | ! |
| 24 | 957.1601 | 954.6148 | 151.4487 | 2.5453 | 400.7 | 0.00635 | 1 1 1 | 0.000 |
| 24 | JJ / . 1001 | )J4.0140 | 131.4407 | 2.3433 | 400.7 | 0.00633 | 1 1 | 1 0.000 |

Sum of Residuals 0
Sum of Squared Residuals 3853369
Predicted Residual SS (PRESS) 5032971

----- SUMMARY REPORT -----Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=Vz\_F

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F
Square

Numerator 2 81235 0.44 0.6481

Denominator 21 183494

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1AUCT

Number of Observations Read 24 Number of Observations Used 24

## Analysis of Variance

DF Sum of Mean F Value Pr > F Source

Squares Square

Model 2 0.30708 0.15354 0.89 0.4272

21 3.63967 0.17332

Corrected Total 23 3.94675

Root MSE 0.41631 R-Square 0.0778 Dependent Mean 7.49304 Adj R-Sq -0.0100

Coeff Var 5.55601

| | | | arameter r | DCIMACC | 2 | |
|---|---|---|---|---|---|---|
| Variable | DF F | Parameter | Standard t | Value F | r > t | 95% |
| | : | Estimate | Error | | | Confidence |
| | | | | | | Limits |
| Intercept | 1 | 7.36860 | 0.14719 | 50.06 | <.0001 | 7.06251 7.67470 |
| GrpA | 1 | 0.09961 | 0.20816 | 0.48 | 0.6372 | -0.33328 0.53249 |
| GrpB | 1 | 0.27371 | 0.20816 | 1.31 | 0.2027 | -0.15917 0.70660 |

# Regression Analysis of Group Child-Pugh Classification at Baseline ------ SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1AUCT

## Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 7.1142 | 7.4682 | 0.1472 | -0.3540 | 0.389 | -0.909 | * | | 0.039 |
| 2 | 7.3961 | 7.4682 | 0.1472 | -0.0721 | 0.389 | -0.185 | | | 0.002 |
| 3 | 6.8861 | 7.4682 | 0.1472 | -0.5821 | 0.389 | -1.495 | ** | | 0.106 |
| 4 | 7.6107 | 7.4682 | 0.1472 | 0.1425 | 0.389 | 0.366 | | | 0.006 |
| 5 | 7.7018 | 7.4682 | 0.1472 | 0.2336 | 0.389 | 0.600 | | * | 0.017 |
| 6 | 7.3802 | 7.4682 | 0.1472 | -0.0880 | 0.389 | -0.226 | | | 0.002 |
| 7 | 7.5766 | 7.4682 | 0.1472 | 0.1084 | 0.389 | 0.278 | | | 0.004 |
| 8 | 8.0799 | 7.4682 | 0.1472 | 0.6117 | 0.389 | 1.571 | | *** | 0.118 |
| 9 | 6.8675 | 7.6423 | 0.1472 | -0.7749 | 0.389 | -1.990 | *** | | 0.189 |
| 10 | 7.5126 | 7.6423 | 0.1472 | -0.1297 | 0.389 | -0.333 | | | 0.005 |
| 11 | 8.1887 | 7.6423 | 0.1472 | 0.5464 | 0.389 | 1.403 | | ** | 0.094 |
| 12 | 7.5410 | 7.6423 | 0.1472 | -0.1013 | 0.389 | -0.260 | | | 0.003 |
| 13 | 7.8972 | 7.6423 | 0.1472 | 0.2549 | 0.389 | 0.654 | | * | 0.020 |
| 14 | 8.0381 | 7.6423 | 0.1472 | 0.3958 | 0.389 | 1.016 | | ** | 0.049 |
| 15 | 6.8784 | 7.6423 | 0.1472 | -0.7639 | 0.389 | -1.962 | *** | | 0.183 |
| 16 | 8.2150 | 7.6423 | 0.1472 | 0.5727 | 0.389 | 1.471 | | ** | 0.103 |
| 17 | 7.5507 | 7.3686 | 0.1472 | 0.1821 | 0.389 | 0.468 | | | 0.010 |
| 18 | 7.5300 | 7.3686 | 0.1472 | 0.1614 | 0.389 | 0.414 | | | 0.008 |
| 19 | 7.5023 | 7.3686 | 0.1472 | 0.1337 | 0.389 | 0.343 | | | 0.006 |
| 20 | 7.4556 | 7.3686 | 0.1472 | 0.0870 | 0.389 | 0.223 | | | 0.002 |
| 21 | 7.0143 | 7.3686 | 0.1472 | -0.3543 | 0.389 | -0.910 | * | | 0.039 |
| 22 | 7.6667 | 7.3686 | 0.1472 | 0.2981 | 0.389 | 0.766 | | * | 0.028 |
| 23 | 6.7872 | 7.3686 | 0.1472 | -0.5815 | 0.389 | -1.493 | ** | | 0.106 |
| 24 | 7.4421 | 7.3686 | 0.1472 | 0.0735 | 0.389 | 0.189 | | | 0.002 |

Sum of Residuals 0
Sum of Squared Residuals 3.63967
Predicted Residual SS (PRESS) 4.75386

----- SUMMARY REPORT -----Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=1AUCT

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 0.15354 0.89 0.4272

Denominator 21 0.17332

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

## Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=lauCinf

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance

DF Sum of Mean F Value Pr > F Source

Squares Square

Model 2 0.36734 0.18367 1.06 0.3639

21 3.63514 0.17310

Corrected Total 23 4.00248

Root MSE 0.41606 R-Square 0.0918 Dependent Mean 7.51869 Adj R-Sq 0.0053

Coeff Var 5.53361

| Variable | DF Parameter | | Standard t | Value Pr > t | | 95% |
|---|---|---|---|---|---|---|
| | Estimate | | Error | Error | | Confidence |
| | | | | | | Limits |
| Intercept | 1 | 7.38275 | 0.14710 | 50.19 | <.0001 | 7.07685 7.68866 |
| GrpA | 1 | 0.10851 | 0.20803 | 0.52 | 0.6074 | -0.32411 0.54113 |
| GrpB | 1 | 0.29930 | 0.20803 | 1.44 | 0.1650 | -0.13332 0.73191 |

## Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=lAUCinf

#### Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 7.1403 | 7.4913 | | | | | * | ı | 0.039 |
| 2 | 7.4226 | 7.4913 | | | 0.389 | | 1 | <br> | 0.001 |
| | | | | | | | 1 | | |
| 3 | 6.9153 | 7.4913 | | | | | ** | | 0.104 |
| 4 | 7.6175 | 7.4913 | | | 0.389 | | | | 0.005 |
| 5 | 7.7251 | 7.4913 | | 0.2338 | 0.389 | | | * | 0.017 |
| 6 | 7.3997 | 7.4913 | 0.1471 | -0.0915 | 0.389 | -0.235 | | | 0.003 |
| 7 | 7.6023 | 7.4913 | 0.1471 | 0.1111 | 0.389 | 0.285 | | | 0.004 |
| 8 | 8.1073 | 7.4913 | 0.1471 | 0.6160 | 0.389 | 1.583 | | *** | 0.119 |
| 9 | 6.9158 | 7.6821 | 0.1471 | -0.7662 | 0.389 | -1.969 | *** | | 0.185 |
| 10 | 7.5340 | 7.6821 | 0.1471 | -0.1481 | 0.389 | -0.380 | | | 0.007 |
| 11 | 8.2456 | 7.6821 | 0.1471 | 0.5636 | 0.389 | 1.448 | | ** | 0.100 |
| 12 | 7.6062 | 7.6821 | 0.1471 | -0.0759 | 0.389 | -0.195 | | | 0.002 |
| 13 | 7.9305 | 7.6821 | 0.1471 | 0.2484 | 0.389 | 0.638 | İ | * | 0.019 |
| 14 | 8.0808 | 7.6821 | 0.1471 | 0.3988 | 0.389 | 1.025 | İ | ** | 0.050 |
| 15 | 6.8940 | 7.6821 | 0.1471 | -0.7880 | 0.389 | -2.025 | **** | | 0.195 |
| 16 | 8.2495 | 7.6821 | 0.1471 | 0.5674 | 0.389 | 1.458 | İ | ** | 0.101 |
| 17 | 7.5616 | 7.3828 | 0.1471 | 0.1789 | 0.389 | 0.460 | | | 0.010 |
| 18 | 7.5339 | 7.3828 | 0.1471 | 0.1511 | 0.389 | 0.388 | İ | | 0.007 |
| 19 | 7.5129 | 7.3828 | 0.1471 | 0.1302 | 0.389 | 0.334 | İ | | 0.005 |
| 20 | 7.4773 | 7.3828 | 0.1471 | 0.0945 | 0.389 | 0.243 | į i | İ | 0.003 |
| 21 | 7.0311 | 7.3828 | 0.1471 | -0.3517 | 0.389 | -0.904 | * | i<br>İ | 0.039 |
| 22 | 7.6717 | 7.3828 | 0.1471 | 0.2890 | 0.389 | 0.742 | i | * | 0.026 |
| 23 | 6.8206 | 7.3828 | | | 0.389 | | ** | | 0.099 |
| 24 | 7.4529 | 7.3828 | | 0.0702 | 0.389 | | j | | 0.002 |

Sum of Residuals 0 Sum of Squared Residuals 3.63514 Predicted Residual SS (PRESS) 4.74794
CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=lauCinf

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 0.18367 1.06 0.3639

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=1CLF

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

Model 2 0.36734 0.18367 1.06 0.3639

21 3.63514 0.17310

Corrected Total 23 4.00248

Root MSE 0.41606 R-Square 0.0918 Dependent Mean 4.68738 Adj R-Sq 0.0053

Coeff Var 8.87606

| Variable | DF : | Parameter | Standard t | Value 1 | Pr > t | 95% |
|---|---|---|---|---|---|---|
| | Estimate | | Error | | | Confidence |
| | | | | | | Limits |
| Intercept | 1 | 4.82332 | 0.14710 | 32.79 | <.0001 | 4.51741 5.12923 |
| GrpA | 1 | -0.10851 | 0.20803 | -0.52 | 0.6074 | -0.54113 0.32411 |
| GrpB | 1 | -0.29930 | 0.20803 | -1.44 | 0.1650 | -0.73191 0.13332 |

# Regression Analysis of Group Child-Pugh Classification at Baseline ------ SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1CLF

# Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 5.0657 | 4.7148 | 0.1471 | 0.3509 | 0.389 | 0.902 | | * | 0.039 |
| 2 | 4.7835 | 4.7148 | 0.1471 | 0.0687 | 0.389 | 0.177 | | | 0.001 |
| 3 | 5.2907 | 4.7148 | 0.1471 | 0.5759 | 0.389 | 1.480 | | ** | 0.104 |
| 4 | 4.5886 | 4.7148 | 0.1471 | -0.1262 | 0.389 | -0.324 | | | 0.005 |
| 5 | 4.4810 | 4.7148 | 0.1471 | -0.2338 | 0.389 | -0.601 | * | | 0.017 |
| 6 | 4.8064 | 4.7148 | 0.1471 | 0.0915 | 0.389 | 0.235 | | | 0.003 |
| 7 | 4.6037 | 4.7148 | 0.1471 | -0.1111 | 0.389 | -0.285 | | | 0.004 |
| 8 | 4.0988 | 4.7148 | 0.1471 | -0.6160 | 0.389 | -1.583 | *** | | 0.119 |
| 9 | 5.2902 | 4.5240 | 0.1471 | 0.7662 | 0.389 | 1.969 | | *** | 0.185 |
| 10 | 4.6721 | 4.5240 | 0.1471 | 0.1481 | 0.389 | 0.380 | | | 0.007 |
| 11 | 3.9604 | 4.5240 | 0.1471 | -0.5636 | 0.389 | -1.448 | ** | | 0.100 |
| 12 | 4.5999 | 4.5240 | 0.1471 | 0.0759 | 0.389 | 0.195 | | | 0.002 |
| 13 | 4.2756 | 4.5240 | 0.1471 | -0.2484 | 0.389 | -0.638 | * | | 0.019 |
| 14 | 4.1253 | 4.5240 | 0.1471 | -0.3988 | 0.389 | -1.025 | ** | | 0.050 |
| 15 | 5.3120 | 4.5240 | 0.1471 | 0.7880 | 0.389 | 2.025 | | **** | 0.195 |
| 16 | 3.9566 | 4.5240 | 0.1471 | -0.5674 | 0.389 | -1.458 | ** | | 0.101 |
| 17 | 4.6445 | 4.8233 | 0.1471 | -0.1789 | 0.389 | -0.460 | | | 0.010 |
| 18 | 4.6722 | 4.8233 | 0.1471 | -0.1511 | 0.389 | -0.388 | | | 0.007 |
| 19 | 4.6932 | 4.8233 | 0.1471 | -0.1302 | 0.389 | -0.334 | | | 0.005 |
| 20 | 4.7288 | 4.8233 | 0.1471 | -0.0945 | 0.389 | -0.243 | | | 0.003 |
| 21 | 5.1750 | 4.8233 | 0.1471 | 0.3517 | 0.389 | 0.904 | | * | 0.039 |
| 22 | 4.5344 | 4.8233 | 0.1471 | -0.2890 | 0.389 | -0.742 | * | | 0.026 |
| 23 | 5.3855 | 4.8233 | 0.1471 | 0.5621 | 0.389 | 1.444 | | ** | 0.099 |
| 24 | 4.7532 | 4.8233 | 0.1471 | -0.0702 | 0.389 | -0.180 | | | 0.002 |

Sum of Residuals 0
Sum of Squared Residuals 3.63514
Predicted Residual SS (PRESS) 4.74794

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=1CLF

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 0.18367 1.06 0.3639

### Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure
Model: MODEL1
Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1Cmax

Number of Observations Read 24 Number of Observations Used 24

# Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

Model 2 0.33702 0.16851 1.03 0.3737

Error 21 3.42932 0.16330

Corrected Total 23 3.76634

Root MSE 0.40410 R-Square 0.0895 Dependent Mean 5.54805 Adj R-Sq 0.0028

Coeff Var 7.28373

| Variable DF Parameter | | Parameter: | Standard t | Value F | r > t | 95% | |
|---|---|---|---|---|---|---|---|
| | | Estimate | | Error | | | Confidence |
| | | | | | | | Limits |
| | Intercept | 1 | 5.39500 | 0.14287 | 37.76 | <.0001 | 5.09788 5.69212 |
| | GrpA | 1 | 0.17046 | 0.20205 | 0.84 | 0.4084 | -0.24973 0.59065 |
| | GrpB | 1 | 0.28870 | 0.20205 | 1.43 | 0.1678 | -0.13149 0.70889 |

# 

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

# Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1Cmax

### Output Statistics

| 01 | D | D 22 2 | Outp | | Ct J D | Q+ | 0 1 | 0 1 0 | G = -1-1 = |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Variable | | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 5.0689 | 5.5655 | 0.1429 | -0.4966 | 0.378 | -1.314 | ** | | 0.082 |
| 2 | 5.8579 | 5.5655 | 0.1429 | 0.2925 | 0.378 | 0.774 | | * | 0.029 |
| 3 | 4.8283 | 5.5655 | 0.1429 | -0.7371 | 0.378 | -1.950 | *** | | 0.181 |
| 4 | 6.2500 | 5.5655 | 0.1429 | 0.6845 | 0.378 | 1.811 | | *** | 0.156 |
| 5 | 5.5413 | 5.5655 | 0.1429 | -0.0242 | 0.378 | -0.0640 | | | 0.000 |
| 6 | 5.5530 | 5.5655 | 0.1429 | -0.0125 | 0.378 | -0.0331 | | | 0.000 |
| 7 | 5.3936 | 5.5655 | 0.1429 | -0.1718 | 0.378 | -0.455 | | | 0.010 |
| 8 | 6.0307 | 5.5655 | 0.1429 | 0.4652 | 0.378 | 1.231 | | ** | 0.072 |
| 9 | 5.3327 | 5.6837 | 0.1429 | -0.3510 | 0.378 | -0.929 | * | | 0.041 |
| 10 | 5.5568 | 5.6837 | 0.1429 | -0.1269 | 0.378 | -0.336 | | | 0.005 |
| 11 | 5.9610 | 5.6837 | 0.1429 | 0.2773 | 0.378 | 0.734 | | * | 0.026 |
| 12 | 5.3982 | 5.6837 | 0.1429 | -0.2855 | 0.378 | -0.755 | * | | 0.027 |
| 13 | 5.8833 | 5.6837 | 0.1429 | 0.1996 | 0.378 | 0.528 | | * | 0.013 |
| 14 | 6.0379 | 5.6837 | 0.1429 | 0.3542 | 0.378 | 0.937 | | * | 0.042 |
| 15 | 4.9628 | 5.6837 | 0.1429 | -0.7209 | 0.378 | -1.907 | *** | | 0.173 |
| 16 | 6.3368 | 5.6837 | 0.1429 | 0.6531 | 0.378 | 1.728 | | *** | 0.142 |
| 17 | 5.2933 | 5.3950 | 0.1429 | -0.1017 | 0.378 | -0.269 | | | 0.003 |
| 18 | 5.7268 | 5.3950 | 0.1429 | 0.3318 | 0.378 | 0.878 | | * | 0.037 |
| 19 | 5.3753 | 5.3950 | 0.1429 | -0.0197 | 0.378 | -0.0522 | | | 0.000 |
| 20 | 5.5984 | 5.3950 | 0.1429 | 0.2034 | 0.378 | 0.538 | | * | 0.014 |
| 21 | 5.2417 | 5.3950 | 0.1429 | -0.1533 | 0.378 | -0.405 | | | 0.008 |
| 22 | 5.6630 | 5.3950 | 0.1429 | 0.2680 | 0.378 | 0.709 | | * | 0.024 |
| 23 | 5.0039 | 5.3950 | 0.1429 | -0.3911 | 0.378 | -1.035 | ** | | 0.051 |
| 24 | 5.2575 | 5.3950 | 0.1429 | -0.1375 | 0.378 | -0.364 | | | 0.006 |
| 24 | 3.23/3 | 5.5550 | 0.1427 | 0.13/3 | 0.570 | 0.304 | 1 | I | |

Sum of Residuals 0 Sum of Squared Residuals 3.42932 Predicted Residual SS (PRESS) 4.47911

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=1Cmax

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 0.16851 1.03 0.3737

# ----- SUMMARY REPORT -----

Algorithme Pharma

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

### Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1LambdaZ

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

Model 2 0.78760 0.39380 10.10 0.0008

21 0.81910 0.03900

Corrected Total 23 1.60669

Root MSE 0.19750 R-Square 0.4902 Dependent Mean -2.17680 Adj R-Sq 0.4416

Coeff Var -9.07279

| Variable | DF Parameter | Standard t | Value Pr | c > t | 95% |
|---|---|---|---|---|---|
| | Estimate | Error | | | Confidence |
| | | | | | Limits |
| Intercept | 1 -1.99319 | 0.06983 - | -28.55 | <.0001 | -2.13840 -1.84798 |
| GrpA | 1 -0.12067 | 0.09875 | -1.22 | 0.2353 | -0.32603 0.08469 |
| GrpB | 1 -0.43014 | 0.09875 | -4.36 | 0.0003 | -0.63549 -0.22478 |

# Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=lLambdaZ

### Output Statistics

| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | -2.3034 | -2.1139 | 0.0698 | -0.1895 | 0.185 | -1.026 | ** | | 0.050 |
| 2 | -2.4392 | -2.1139 | 0.0698 | -0.3253 | 0.185 | -1.761 | *** | | 0.148 |
| 3 | -1.8463 | -2.1139 | 0.0698 | 0.2675 | 0.185 | 1.448 | | ** | 0.100 |
| 4 | -1.6405 | -2.1139 | 0.0698 | 0.4734 | 0.185 | 2.562 | | **** | 0.313 |
| 5 | -2.2706 | -2.1139 | 0.0698 | -0.1568 | 0.185 | -0.849 | * | | 0.034 |
| 6 | -1.8062 | -2.1139 | 0.0698 | 0.3077 | 0.185 | 1.665 | | *** | 0.132 |
| 7 | -2.3217 | -2.1139 | 0.0698 | -0.2079 | 0.185 | -1.125 | ** | | 0.060 |
| 8 | -2.2829 | -2.1139 | 0.0698 | -0.1691 | 0.185 | -0.915 | * | | 0.040 |
| 9 | -2.2587 | -2.4233 | 0.0698 | 0.1646 | 0.185 | 0.891 | | * | 0.038 |
| 10 | -2.3614 | -2.4233 | 0.0698 | 0.0619 | 0.185 | 0.335 | | | 0.005 |
| 11 | -2.5551 | -2.4233 | 0.0698 | -0.1318 | 0.185 | -0.713 | * | | 0.024 |
| 12 | -2.6217 | -2.4233 | 0.0698 | -0.1984 | 0.185 | -1.074 | ** | | 0.055 |
| 13 | -2.4174 | -2.4233 | 0.0698 | 0.005937 | 0.185 | 0.0321 | | | 0.000 |
| 14 | -2.5264 | -2.4233 | 0.0698 | -0.1031 | 0.185 | -0.558 | * | | 0.015 |
| 15 | -2.2508 | -2.4233 | 0.0698 | 0.1726 | 0.185 | 0.934 | | * | 0.042 |
| 16 | -2.3951 | -2.4233 | 0.0698 | 0.0282 | 0.185 | 0.153 | | | 0.001 |
| 17 | -2.0608 | -1.9932 | 0.0698 | -0.0676 | 0.185 | -0.366 | | | 0.006 |
| 18 | -1.8844 | -1.9932 | 0.0698 | 0.1088 | 0.185 | 0.589 | | * | 0.017 |
| 19 | -2.0951 | -1.9932 | 0.0698 | -0.1019 | 0.185 | -0.552 | * | | 0.014 |
| 20 | -1.9182 | -1.9932 | 0.0698 | 0.0750 | 0.185 | 0.406 | | | 0.008 |
| 21 | -1.8884 | -1.9932 | 0.0698 | 0.1048 | 0.185 | 0.567 | | * | 0.015 |
| 22 | -1.9465 | -1.9932 | 0.0698 | 0.0467 | 0.185 | 0.253 | | | 0.003 |
| 23 | -2.0413 | -1.9932 | 0.0698 | -0.0481 | 0.185 | -0.261 | | | 0.003 |
| 24 | -2.1108 | -1.9932 | 0.0698 | -0.1176 | 0.185 | -0.637 | * | | 0.019 |

Sum of Residuals 0 Sum of Squared Residuals 0.81910 Predicted Residual SS (PRESS) 1.06984 Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=lLambdaZ

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 2 0.39380 10.10 0.0008

### Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

NAME OF FORMER VARIABLE=1Vz F

Number of Observations Read 24 Number of Observations Used 24

Analysis of Variance

Source DF Sum of Mean F Value Pr > F

Squares Square

Model 2 0.08360 0.04180 0.26 0.7713

21 3.33827 0.15897

Corrected Total 23 3.42187

Root MSE 0.39870 R-Square 0.0244 Dependent Mean 6.86418 Adj R-Sq -0.0685

Coeff Var 5.80848

| Variable | DF F | arameter | Standard t | Value P | r > t | 95% |
|---|---|---|---|---|---|---|
| | Estimate | | Error | | | Confidence |
| | | | | | | Limits |
| Intercept | 1 | 6.81651 | 0.14096 | 48.36 | <.0001 | 6.52336 7.10966 |
| GrpA | 1 | 0.01216 | 0.19935 | 0.06 | 0.9519 | -0.40242 0.42674 |
| GrpB | 1 | 0.13084 | 0.19935 | 0.66 | 0.5187 | -0.28374 0.54541 |

# Regression Analysis of Group Child-Pugh Classification at Baseline ----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### NAME OF FORMER VARIABLE=1Vz F

# Output Statistics

| Obs | Dependent<br>Variable | | Std Error Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 7.3691 | 6.8287 | 0.1410 | 0.5405 | 0.373 | 1.449 | | ** | 0.100 |
| 2 | 7.2227 | 6.8287 | 0.1410 | 0.3940 | 0.373 | 1.057 | | ** | 0.053 |
| 3 | 7.1371 | 6.8287 | 0.1410 | 0.3084 | 0.373 | 0.827 | | * | 0.033 |
| 4 | 6.2291 | 6.8287 | 0.1410 | -0.5996 | 0.373 | -1.608 | *** | | 0.123 |
| 5 | 6.7516 | 6.8287 | 0.1410 | -0.0770 | 0.373 | -0.207 | | | 0.002 |
| 6 | 6.6126 | 6.8287 | 0.1410 | -0.2161 | 0.373 | -0.579 | * | | 0.016 |
| 7 | 6.9255 | 6.8287 | 0.1410 | 0.0968 | 0.373 | 0.260 | | | 0.003 |
| 8 | 6.3818 | 6.8287 | 0.1410 | -0.4469 | 0.373 | -1.198 | ** | | 0.068 |
| 9 | 7.5490 | 6.9474 | 0.1410 | 0.6016 | 0.373 | 1.613 | | *** | 0.124 |
| 10 | 7.0335 | 6.9474 | 0.1410 | 0.0862 | 0.373 | 0.231 | | | 0.003 |
| 11 | 6.5155 | 6.9474 | 0.1410 | -0.4318 | 0.373 | -1.158 | ** | | 0.064 |
| 12 | 7.2216 | 6.9474 | 0.1410 | 0.2743 | 0.373 | 0.735 | | * | 0.026 |
| 13 | 6.6930 | 6.9474 | 0.1410 | -0.2543 | 0.373 | -0.682 | * | | 0.022 |
| 14 | 6.6517 | 6.9474 | 0.1410 | -0.2957 | 0.373 | -0.793 | * | | 0.030 |
| 15 | 7.5628 | 6.9474 | 0.1410 | 0.6154 | 0.373 | 1.650 | | *** | 0.130 |
| 16 | 6.3517 | 6.9474 | 0.1410 | -0.5956 | 0.373 | -1.597 | *** | | 0.121 |
| 17 | 6.7052 | 6.8165 | 0.1410 | -0.1113 | 0.373 | -0.298 | | | 0.004 |
| 18 | 6.5566 | 6.8165 | 0.1410 | -0.2600 | 0.373 | -0.697 | * | | 0.023 |
| 19 | 6.7883 | 6.8165 | 0.1410 | -0.0282 | 0.373 | -0.0756 | | | 0.000 |
| 20 | 6.6470 | 6.8165 | 0.1410 | -0.1695 | 0.373 | -0.455 | | | 0.010 |
| 21 | 7.0634 | 6.8165 | 0.1410 | 0.2469 | 0.373 | 0.662 | | * | 0.021 |
| 22 | 6.4808 | 6.8165 | 0.1410 | -0.3357 | 0.373 | -0.900 | * | | 0.039 |
| 23 | 7.4268 | 6.8165 | 0.1410 | 0.6103 | 0.373 | 1.636 | | *** | 0.128 |
| 24 | 6.8640 | 6.8165 | 0.1410 | 0.0475 | 0.373 | 0.127 | | | 0.001 |

Sum of Residuals 0 Sum of Squared Residuals 3.33827 Predicted Residual SS (PRESS) 4.36019

CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

Regression Analysis of Group Child-Pugh Classification at Baseline

----- SUMMARY REPORT -----

The REG Procedure Model: MODEL1

NAME OF FORMER VARIABLE=1Vz\_F

Test test FunctionGroup Results for Dependent Variable Value

Source DF Mean F Value Pr > F Square

Numerator 

Algorithme Pharma

#### CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

# NON-PARAMETRIC TEST OF FIXED EFFECT for Tmax parameter ----- SUMMARY REPORT -----

#### The NPAR1WAY Procedure

Wilcoxon Scores (Rank Sums) for Variable Value Classified by Variable FunctionGroup

N Sum of Expected Std Dev Mean Scores Under H0 Under H0 Score FunctionGroup 2 8 38.50 68.0 9.465728 4.81250 3 8 97.50 68.0 9.465728 12.18750

Average scores were used for ties.

Wilcoxon Two-Sample Test

Statistic 38.5000

Normal Approximation

-3.0637 One-Sided Pr < Z 0.0011 Two-Sided Pr > |Z|0.0022

t Approximation

One-Sided Pr < Z 0.0039 Two-Sided Pr > |Z| 0.0079

Z includes a continuity correction of 0.5.

Kruskal-Wallis Test

Chi-Square 9.7126 1 DF Pr > Chi-Square 0.0018

Hodges-Lehmann Estimation Location Shift (2 - 3) -1.2500

90% Interval Asymptotic Confidence Midpoint Standard Error

Limits

Asymptotic (Moses) -2.0000 -0.5333 -1.2667

Exact -2.0000 -0.7500 -1.3750

# NON-PARAMETRIC TEST OF FIXED EFFECT for Tmax parameter ----- SUMMARY REPORT -----

#### The NPAR1WAY Procedure

Wilcoxon Scores (Rank Sums) for Variable Value Classified by Variable FunctionGroup

N Sum of Expected Std Dev Mean Scores Under H0 Under H0 Score FunctionGroup 1 8 52.50 68.0 9.402127 6.56250 8 83.50 68.0 9.402127 10.43750 3

Average scores were used for ties.

Wilcoxon Two-Sample Test

Statistic 52.5000

Normal Approximation

-1.5954 One-Sided Pr < Z 0.0553 Two-Sided Pr > |Z|0.1106

t Approximation

One-Sided Pr < Z 0.0657 Two-Sided Pr > |Z| 0.1315

Z includes a continuity correction of 0.5.

Kruskal-Wallis Test

Chi-Square 2.7178 1 DF Pr > Chi-Square 0.0992

Hodges-Lehmann Estimation Location Shift (1 - 3) -1.0000

90% Interval Asymptotic Confidence Midpoint Standard Error

Limits

Asymptotic (Moses) -1.7500 0.0000 -0.8750 Exact -1.7500 0.0000 -0.8750

Algorithme Pharma

#### CUD-P9-453: Effect of Hepatic Impairment on Pharmacokinetics of Lasmiditan

# NON-PARAMETRIC TEST OF FIXED EFFECT for Tmax parameter ----- SUMMARY REPORT -----

#### The NPAR1WAY Procedure

Wilcoxon Scores (Rank Sums) for Variable Value Classified by Variable FunctionGroup

N Sum of Expected Std Dev Mean Scores Under H0 Under H0 Score FunctionGroup 8 81.0 68.0 9.423375 10.1250 8 55.0 68.0 9.423375 6.8750 2

Average scores were used for ties.

Wilcoxon Two-Sample Test

Statistic 81.0000 Normal Approximation 1.3265 One-Sided Pr > Z 0.0923 Two-Sided Pr > |Z| 0.1847 t Approximation One-Sided Pr > Z 0.1023 Two-Sided Pr > |Z| 0.2045

Z includes a continuity correction of 0.5.

Kruskal-Wallis Test

Chi-Square 1.9032 DF 1 Pr > Chi-Square 0.1677

Hodges-Lehmann Estimation

Location Shift (1 - 2) 0.5000
90% Interval Asymptotic Confidence Midpoint Standard Error Limits

Asymptotic (Moses) -0.2500 1.2500 0.5000 Exact 0.0000 1.2500 0.6250